CLINICAL TRIAL: NCT04575597
Title: A Phase 2/3, Randomized, Placebo-Controlled, Double-Blind Clinical Study to Evaluate the Efficacy, Safety, and Pharmacokinetics of MK-4482 in Non-Hospitalized Adults With COVID-19.
Brief Title: Efficacy and Safety of Molnupiravir (MK-4482) in Non-Hospitalized Adult Participants With COVID-19 (MK-4482-002)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4482-002; MK-4482-002 (Other: Merck); PHRR201209-003186 (Registry Identifier: PHRR); jRCT2031210148 (Registry Identifier: jRCT); 2020-003368-24 (EudraCT Number)
Record Dates: First submitted 2020-09-30; First posted 2020-10-05 (Actual); Results first posted 2023-06-28 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-05

CONDITIONS: Coronavirus Disease (COVID-19)
MeSH Terms: conditions — COVID-19 | interventions — molnupiravir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Part 1: Molnupiravir 200 mg (Experimental): 200 mg molnupiravir administered orally every 12 hours for 5 days (10 doses total)
  Interventions: Drug: Molnupiravir
- Part 1: Molnupiravir 400 mg (Experimental): 400 mg molnupiravir administered orally every 12 hours for 5 days (10 doses total)
  Interventions: Drug: Molnupiravir
- Part 1: Molnupiravir 800 mg (Experimental): 800 mg molnupiravir administered orally every 12 hours for 5 days (10 doses total)
  Interventions: Drug: Molnupiravir
- Part 1: Placebo (Placebo Comparator): Placebo matching molnupiravir administered orally every 12 hours for 5 days (10 doses total)
  Interventions: Drug: Placebo
- Part 2: Molnupiravir 800 mg (Experimental): 800 mg Molnupiravir (dose to be selected) administered orally every 12 hours for 5 days (10 doses total)
  Interventions: Drug: Molnupiravir
- Part 2: Placebo (Placebo Comparator): Placebo matching molnupiravir administered orally every 12 hours for 5 days (10 doses total)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Molnupiravir — Molnupiravir administered orally in capsule form every 12 hours for 5 days (10 doses total)
  Other Names: MK-4482
  Arms: Part 1: Molnupiravir 200 mg; Part 1: Molnupiravir 400 mg; Part 1: Molnupiravir 800 mg; Part 2: Molnupiravir 800 mg
Drug: Placebo — Placebo matching molnupiravir administered orally in capsule form every 12 hours for 5 days (10 doses total)
  Arms: Part 1: Placebo; Part 2: Placebo

SUMMARY:
This study aims to evaluate the safety, tolerability and efficacy of molnupiravir (MK-4482) compared to placebo. The primary hypothesis is that molnupiravir is superior to placebo as assessed by the percentage of participants who are hospitalized and/or die through Day 29

ELIGIBILITY:
Inclusion Criteria:

* Has documentation of laboratory confirmed severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection with sample collection ≤5 days prior to the day of randomization. PCR is the preferred method; however with evolving approaches to laboratory confirmation of SARS-CoV-2 infection, other molecular or antigen tests that detect viral ribonucleic acid (RNA) or protein are allowed if authorized for use in the country. Serological tests that detect host antibodies generated in response to recent or prior infection are not allowed.
* Had initial onset of signs/symptoms attributable to COVID-19 for ≤5 days prior to the day of randomization and at least 1 of the following sign/symptom attributable to COVID-19 on the day of randomization.
* Has mild or moderate COVID-19.
* Has at least 1 characteristic or underlying medical condition associated with an increased risk of severe illness from COVID-19.
* Males agree to the following during the intervention period and for at least 4 days after the last dose of study intervention: Either abstain from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis) and agree to remain abstinent; or must agree to use contraception.
* Females are not pregnant or breastfeeding, and at least one of the following conditions applies: Is not a woman of child bearing potential (WOCBP); or is a WOCBP and using a contraceptive method that is highly effective (a low user dependency method OR a user dependent method in combination with barrier method), or be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long-term and persistent basis) for at least 4 days after the last dose of study intervention; a WOCBP must have a negative highly sensitive pregnancy test (urine or serum test is required) within 24 hours before the first dose of study intervention.

Exclusion Criteria:

* Is currently hospitalized or is expected to need hospitalization for COVID-19 within 48 hours of randomization.
* Is on dialysis or has reduced estimated glomerular filtration rate (eGFR) <30 mL/min/1.73m^2 by the Modification of Diet in Renal Disease (MDRD) equation.
* Has any of the following conditions: human immunodeficiency virus (HIV) with a recent viral load >50 copies/mL (regardless of CD4 count) or an AIDS-defining illness in the past 6 months, participants with HIV may only be enrolled if on a stable antiretroviral therapy regimen; a neutrophilic granulocyte absolute count <500/mm^3.
* Has a history of hepatitis B virus (HBV) or hepatitis C virus (HCV) with cirrhosis, end-stage liver disease, hepatocellular carcinoma, aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) >3X upper limit of normal at screening.
* Has a platelet count <100,000/μL or received a platelet transfusion in the 5 days prior to randomization.
* Is taking or is anticipated to require any prohibited therapies.
* Is unwilling to abstain from participating in another interventional clinical study through Day 29 with an investigational compound or device, including those for COVID-19 therapeutics.
* Has hypersensitivity or other contraindication to any of the components of the study interventions as determined by the investigator.
* Has any condition for which, in the opinion of the investigator, participation would not be in the best interest of the participant or that could prevent, limit, or confound the protocol-specified assessments including but not limited to: participants who are not expected to survive longer than 48 hours after randomization, or participants with a recent history of mechanical ventilation, or participants with conditions that could limit gastrointestinal absorption of capsule contents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1735 (Actual)
Dates: Start 2020-10-19 (Actual); Primary Completion 2022-05-05 (Actual); Study Completion 2022-05-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (173):
- United States (32):
  - Phoenix Medical Group ( Site 1822), Peoria, Arizona
  - Ruane Clinical Research Group, Inc. ( Site 2406), Los Angeles, California
  - Men's Health Foundation ( Site 1820), Los Angeles, California
  - Carbon Health Technologies Inc ( Site 2505), North Hollywood, California
  - UC Davis Medical Center ( Site 1833), Sacramento, California
  - Emerson Clinical Research Institute ( Site 1828), Washington D.C., District of Columbia
  - JEM Research Institute ( Site 2508), Atlantis, Florida
  - Midway Immunology and Research Center ( Site 1837), Ft. Pierce, Florida
  - Indago Research & Health Center, Inc ( Site 1809), Hialeah, Florida
  - Advanced Research For Health Improvement LLC ( Site 1816), Immokalee, Florida
  - Advanced Medical Research, LLC ( Site 1864), Miami, Florida
  - Advanced Research For Health Improvement LLC ( Site 1813), Naples, Florida
  - Bliss Healthcare Services ( Site 1847), Orlando, Florida
  - Javara Inc. ( Site 1869), Albany, Georgia
  - IACT Health ( Site 1818), Columbus, Georgia
  - Javara Inc. ( Site 1868), Fayetteville, Georgia
  - Loretto Hospital ( Site 1886), Chicago, Illinois
  - Jadestone Clinical Research, LLC ( Site 2502), Laurel, Maryland
  - Michigan Center of Medical Research ( Site 2500), Farmington Hills, Michigan
  - University of Nebraska Medical Center ( Site 2414), Omaha, Nebraska
  - Amici Clinical Research LLC ( Site 2507), Raritan, New Jersey
  - University of New Mexico, Health Sciences Center ( Site 1819), Albuquerque, New Mexico
  - AXCES Research Group ( Site 2418), Santa Fe, New Mexico
  - Saint Hope Foundation, Inc. ( Site 1830), Bellaire, Texas
  - The Crofoot Research Center, Inc. ( Site 1812), Houston, Texas
  - Javara Inc. ( Site 1866), Sugar Land, Texas
  - Clinical Research Partners, LLC. ( Site 2503), Richmond, Virginia
  - Swedish Medical Center First Hill ( Site 1807), Seattle, Washington
  - Fred Hutchinson Cancer Center ( Site 1829), Seattle, Washington
  - Multicare Health System ( Site 1811), Spokane, Washington
  - Multicare Health System ( Site 1814), University Place, Washington
  - Medical College Of Wisconsin ( Site 2510), Milwaukee, Wisconsin
- Argentina (2):
  - Clinica Independencia ( Site 3400), Vicente López, Buenos Aires
  - Instituto Medico de la Fundacion Estudios Clinicos ( Site 3401), Rosario, Santa Fe Province
- Brazil (7):
  - Chronos Pesquisa Clínica ( Site 0155), Brasília, Federal District
  - Santa Casa de Misericordia de Belo Horizonte ( Site 0150), Belo Horizonte, Minas Gerais
  - Hospital de Clinicas da Universidade Federal do Parana ( Site 0154), Curitiba, Paraná
  - Hospital Tacchini ( Site 0157), Bento Gonçalves, Rio Grande do Sul
  - FUNFARME Hospital de Base Centro Integrado de Pesquisa ( Site 0151), São José do Rio Preto, São Paulo
  - Instituto de Infectologia Emilio Ribas ( Site 0153), São Paulo
  - Centro de Pesquisa Clinica II - ICHC - FMUSP ( Site 0152), São Paulo
- Canada (4):
  - Hamilton Medical Research Group ( Site 0207), Hamilton, Ontario
  - University Health Network - Toronto General Hospital ( Site 0201), Toronto, Ontario
  - Centre Hospitalier de l Universite de Montreal - CHUM ( Site 0200), Montreal, Quebec
  - McGill University Health Centre ( Site 0204), Montreal, Quebec
- Chile (7):
  - Servicios Medicos Urumed ( Site 0307), Rancagua, Lbtdr Gen Bernardo O Higgins
  - Clinical Research Chile SpA ( Site 0308), Valdivia, Los Ríos Region
  - Clinica Universidad de los Andes ( Site 0302), Santiago, Region M. de Santiago
  - Fundacion Arturo Lopez Perez ( Site 0305), Santiago, Region M. de Santiago
  - Espacio EME ( Site 0304), Santiago, Region M. de Santiago
  - Centro de Investigacion Clinica UC CICUC ( Site 0309), Santiago, Region M. de Santiago
  - Clinica Bicentenario Spa ( Site 0306), Santiago, Region M. de Santiago
- Colombia (10):
  - Hospital Pablo Tobon Uribe ( Site 0405), Medellín, Antioquia
  - Centro Cientifico Asistencial Jose Luis Accini ( Site 0416), Barranquilla, Atlántico
  - Clinica de la Costa Ltda. ( Site 0403), Barranquilla, Atlántico
  - Fundacion Santa Fe de Bogota ( Site 0412), Bogotá, Bogota D.C.
  - Caja de Compensación Familiar CAFAM. Sede Centro de Atención en Salud CAFAM Floresta ( Site 0406), Bogota, Cundinamarca
  - Centro de Atencion e Investigacion Medica CAIMED ( Site 0413), Bogota, Cundinamarca
  - Oncomedica S.A. ( Site 0407), Montería, Departamento de Córdoba
  - Fundacion Cardiovascular de Colombia ( Site 0402), Bucaramanca, Santander Department
  - Fundacion Valle del Lili ( Site 0401), Cali, Valle del Cauca Department
  - Centro Medico Imbanaco de Cali S.A ( Site 0415), Cali, Valle del Cauca Department
- Egypt (5):
  - National Hepatology & Tropical Medicine Research Institute (NHTMRI) ( Site 3300), Cairo, Cairo Governorate
  - Abbassia Chest Hospital ( Site 3340), Cairo, Cairo Governorate
  - Abbassia Fever Hospital ( Site 3330), Cairo, Cairo Governorate
  - Helwan Fever Hospital ( Site 3350), Cairo, Cairo Governorate
  - National Center for allergies and chest ( Site 3320), Giza, Giza Governorate
- France (8):
  - Hopital Bichat Claude Bernard ( Site 0503), Paris, Ain
  - Hopital Saint Joseph ( Site 0513), Marseille, Bouches-du-Rhone
  - Groupe Hospitalier Pellegrin ( Site 0511), Bordeaux, Gironde
  - CHU de la Reunion - Groupe Hospitalier Sud ( Site 0514), Saint-Pierre, La Reunion
  - C.H.U. de Toulouse Hopital Purpan ( Site 0501), Toulouse, Midi-Pyrenees
  - Centre Hospitalier de Tourcoing ( Site 0502), Tourcoing, Nord
  - CHU Hopital Saint Antoine ( Site 0505), Paris
  - Pitie Salpetriere University Hospital-Infectious Disease - Tropical Diseases ( Site 0504), Paris
- Germany (4):
  - Universitaetsklinikum Frankfurt ( Site 2302), Frankfurt A Main, Hesse
  - Universitaetsklinikum Essen ( Site 2305), Essen, North Rhine-Westphalia
  - ZIBP-Zentrum fur Infektiologie Berlin Prenzlauer Berg GmbH ( Site 2301), Berlin
  - ICH Study Center GmbH & Co.KG ( Site 2306), Hamburg
- Guatemala (2):
  - Clínica Médica Especializada en Pediatría e Infectología Pediátrica - Dr. Mario Melgar ( Site 2601), Guatemala City
  - Clinica Privada Dr. Jose Francisco Flores Lopez ( Site 2600), Guatemala City
- Hadassah Medical Center. Ein Kerem ( Site 2100), Jerusalem, Israel
- Italy (11):
  - Asl Napoli 1 Centro ( Site 0610), Naples, Napoli
  - Policlinico S. Orsola-Malpighi ( Site 0604), Bologna
  - IRCCS Ospedale Policlinico San Martino ( Site 0603), Genova
  - Fondazione IRCCS Ca' Granda-Ospedale Maggiore Policlinico ( Site 0606), Milan
  - Ospedale San Raffaele ( Site 0605), Milan
  - ASST Fatebenefratelli-Ospedale Sacco ( Site 0601), Milan
  - Ospedale Niguarda ( Site 0608), Milan
  - AOU Policlinico Paolo Giaccone ( Site 0609), Palermo
  - Istituto Nazionale per Le Malattie Infettive Lazzaro Spallanzani ( Site 0600), Roma
  - Ospedale Amedeo di Savoia, Malattie Infettive ( Site 0602), Torino
  - Azienda Sanitaria Universitaria Friuli Centrale -ASU FC ( Site 0607), Udine
- Japan (3):
  - Chiba Aoba Municipal Hospital ( Site 0702), Chiba
  - Den-en-chofu family clinic ( Site 0701), Tokyo
  - Center Hospital of the National Center for Global Health and Medicine ( Site 0700), Tokyo
- Mexico (11):
  - Hospital Regional de Alta Especialidad del Bajio ( Site 0807), León, Guanajuato
  - Hospital Civil de Guadalajara Fray Antonio Alcalde ( Site 0800), Guadalajara, Jalisco
  - CAIMED México ( Site 0814), Mexico City, Mexico City
  - Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran ( Site 0802), Mexico City, Mexico City
  - Hospital Universitario Dr. Jose Eleuterio Gonzalez ( Site 0803), Monterrey, Nuevo León
  - Centro de Investigacion y Avances Medicos Especializados -CIAME ( Site 0810), Cancún, Quintana Roo
  - Köhler & Milstein Research S.A. de C.V. ( Site 0809), Mérida, Yucatán
  - ICARO Investigaciones en Medicina ( Site 0812), Chihuahua City
  - Oaxaca Site Management Organization S.C. ( Site 0811), Oaxaca City
  - Clinical Research Institute S.C. ( Site 0813), Tlalnepantla
  - Arké SMO S.A de C.V ( Site 0808), Veracruz
- Philippines (2):
  - Lung Center of the Philippines ( Site 0902), Quezon City, National Capital Region
  - Quirino Memorial Medical Center ( Site 0903), Quezon City, National Capital Region
- Poland (4):
  - Krakowskie Centrum Medyczne Sp. z o.o ( Site 1008), Krakow, Lesser Poland Voivodeship
  - Centrum Medyczne Pulawska Sp. z o.o. ( Site 1007), Piaseczno, Masovian Voivodeship
  - Centrum Medyczne MEDYK Sp. z o.o. Sp.k. ( Site 1009), Rzeszów, Podkarpackie Voivodeship
  - NZOZ Centrum Medyczne Szpital Swietej Rodziny ( Site 1006), Lodz, Łódź Voivodeship
- Russia (15):
  - Central Scientific Research Institute of Epidemiology ( Site 1104), Moscow, Moscow
  - Open Joint Stock Company Clinical and Diagnostic Center Euromedservice ( Site 1122), Moscow, Moscow
  - Hadassah Medical LTD ( Site 1124), Moscow, Moscow
  - Central Clinical Hospital with Polyclinic ( Site 1105), Moscow, Moscow
  - City Hospital No.33 of Leninsky ( Site 1127), Nizhny Novgorod, Nizhny Novgorod Oblast
  - City Polyclinic N44 ( Site 1130), Saint Petersburg, Sankt-Peterburg
  - Strategic Medical System LLC ( Site 1114), Saint Petersburg, Sankt-Peterburg
  - St.Petersburg Outpatient Clinic No. 109 ( Site 1119), Saint Petersburg, Sankt-Peterburg
  - SPb SBHI City outpatient clinic 112 ( Site 1128), Saint Petersburg, Sankt-Peterburg
  - Medical Research Institute LLC ( Site 1116), Saint Petersburg, Sankt-Peterburg
  - Limited liability company "Scientific research center Eco-safety" ( Site 1117), Saint Petersburg, Sankt-Peterburg
  - Smorodintsev Research Institute of Influenza ( Site 1129), Saint Petersburg, Sankt-Peterburg
  - SPb SBHI City outpatient clinic 4 ( Site 1131), Saint Petersburg, Sankt-Peterburg
  - Smolensk State Medical University ( Site 1110), Smolensk, Smolensk Oblast
  - Republican Clinical Infectious Hospital n.a. A.F. Agafonov ( Site 1100), Kazan', Tatarstan, Respublika
- South Africa (12):
  - IATROS International ( Site 1212), Bloemfontein, Free State
  - Right To Care Research - Esizayo ( Site 1229), Johannesburg, Gauteng
  - Mzansi Ethical Research Centre ( Site 1225), Mpumalanga, Gauteng
  - Jongaie Research ( Site 1223), Pretoria West, Gauteng
  - Wits Baragwanath Clinical Trial Site ( Site 1214), Soweto, Gauteng
  - Enhancing Care Foundation-DICRS ( Site 1216), Durban, KwaZulu-Natal
  - Limpopo Clinical Research Initiative ( Site 1227), Thabazimbi, Limpopo
  - TREAD Research ( Site 1211), Cape Town, Western Cape
  - Desmond Tutu HIV Foundation Clinical Trial Unit ( Site 1219), Cape Town, Western Cape
  - Be Part Yoluntu Centre ( Site 1218), Paarl, Western Cape
  - Paarl Research Centre ( Site 1228), Paarl, Western Cape
  - Clinical Projects Research Centre ( Site 1215), Worcester, Western Cape
- Spain (9):
  - CAP Centelles ( Site 1308), Centelles, Barcelona
  - Fundacion Hospital Alcorcon de Madrid ( Site 1314), Alcorcón, Madrid
  - Hospital General Universitario Gregorio Maranon ( Site 1302), Madrid, Madrid, Comunidad de
  - CAP Sardenya - Barcelona ( Site 1307), Barcelona
  - Hospital Clinic ( Site 1304), Barcelona
  - Hospital Universitari Germans Trias i Pujol ( Site 1303), Barcelona
  - Hospital Universitario Infanta Leonor ( Site 1310), Madrid
  - Hospital Universitario Ramon y Cajal ( Site 1301), Madrid
  - Hospital Universitario La Paz ( Site 1300), Madrid
- Sweden (3):
  - Karolinska Universitetssjukhuset Solna ( Site 1400), Stockholm, Stockholm County
  - ClinSmart Sweden AB.Uppsala ( Site 1402), Uppsala, Uppsala County
  - Sahlgrenska Universitetssjukhuset Ostra ( Site 1401), Gothenburg, Västra Götaland County
- Taiwan (2):
  - National Taiwan University Hospital ( Site 3100), Taipei
  - Taoyuan General Hospital ( Site 3101), Taoyuan District
- Ukraine (13):
  - Ivano-Frankivsk Regional Clinical Infectious Diseases Hospital ( Site 1605), Ivano-Frankivsk, Ivano-Frankivsk Oblast
  - CNE Central city clinical hospital of Ivano-Frankivsk city council ( Site 1604), Ivano-Frankivsk, Ivano-Frankivsk Oblast
  - MNE Ivano-Frankivsk Regional Phthisiology-Pulmonology Center ( Site 1603), Ivano-Frankivsk, Ivano-Frankivsk Oblast
  - Non profit municipal enterprise City hospital student of Kharkiv city council ( Site 1621), Kharkiv, Kharkivs’ka Oblast’
  - PCNE Kharkiv City polyclinic 9 of the Kharkiv City Council ( Site 1627), Kharkiv, Kharkivs’ka Oblast’
  - Limited Liability Company Medical center Healthy Happy ( Site 1625), Kyiv, Kyivska Oblast
  - LLC "Adonis plus" ( Site 1619), Kyiv, Kyivska Oblast
  - Kyiv railway clinical hospital 2 of Branch Health center ( Site 1602), Kyiv, Kyivska Oblast
  - ARTEM. State Holding Company ( Site 1618), Kyiv, Kyivska Oblast
  - Municipal Noncommercial Enterprise Lviv 4th City Clinical Hospital ( Site 1622), Lviv, Lviv Oblast
  - MNCE -Odesa regional clinical hospital of Odesa regional council ( Site 1626), Odesa, Odesa Oblast
  - Municipal Enterprise Poltava Regional Clinical Infectious Hospital ( Site 1614), Poltava, Poltava Oblast
  - Medical Center Health Clinic ( Site 1623), Vinnytsia, Vinnytsia Oblast
- United Kingdom (6):
  - The Adam Practice ( Site 1708), Poole, Dorset
  - Accellacare South London Quality Research Centre ( Site 1709), Orpington, Kent
  - Royal Free London NHS Foundation Trust ( Site 1700), London, London, City of
  - King's College Hospital ( Site 1707), London, London, City of
  - Layton Medical Centre ( Site 1705), Blackpool
  - Newcastle upon Tyne Hospitals NHS Foundation Trust ( Site 1704), Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Caraco Y, Crofoot GE, Moncada PA, Galustyan AN, Musungaie DB, Payne B, Kovalchuk E, Gonzalez A, Brown ML, Williams-Diaz A, Gao W, Strizki JM, Grobler J, Du J, Assaid CA, Paschke A, Butterton JR, Johnson MG, De Anda C. Phase 2/3 Trial of Molnupiravir for Treatment of Covid-19 in Nonhospitalized Adults. NEJM Evid. 2022 Feb;1(2):EVIDoa2100043. doi: 10.1056/EVIDoa2100043. Epub 2021 Dec 16. PMID 38319179
- [Derived] Johnson MG, Strizki JM, Hilbert DW, Zhang Y, Carmelitano P, Brown ML, Wolf DJ, Paschke A, De Anda CS. Impact of baseline humoral immunity on treatment outcomes with molnupiravir in the MOVe-OUT randomized, controlled trial. Virology. 2026 Jan;613:110710. doi: 10.1016/j.virol.2025.110710. Epub 2025 Oct 9. PMID 41125063
- [Derived] Caraco Y, Johnson MG, Chiarappa JA, Maas BM, Stone JA, Rizk ML, Vesnesky M, Strizki JM, Williams-Diaz A, Brown ML, Carmelitano P, Wan H, Pedley A, Chawla A, Wolf DJ, Grobler JA, Paschke A, De Anda C. Impact of differences between interim and post-interim analysis populations on outcomes of a group sequential trial: Example of the MOVe-OUT study. Clin Trials. 2025 Jun;22(3):312-324. doi: 10.1177/17407745251313925. Epub 2025 Mar 2. PMID 40025641
- [Derived] Strizki JM, Grobler JA, Murgolo N, Fridman A, Johnson MG, Du J, Carmelitano P, Brown ML, Paschke A, De Anda C. Virologic Outcomes with Molnupiravir in Non-hospitalized Adult Patients with COVID-19 from the Randomized, Placebo-Controlled MOVe-OUT Trial. Infect Dis Ther. 2023 Dec;12(12):2725-2743. doi: 10.1007/s40121-023-00891-1. Epub 2023 Nov 23. PMID 37995070
- [Derived] Guan Y, Puenpatom A, Johnson MG, Zhang Y, Zhao Y, Surber J, Weinberg A, Brotons C, Kozlov R, Lopez R, Coetzee K, Santiaguel J, Du J, Williams-Diaz A, Brown M, Paschke A, De Anda C, Norquist JM. Impact of Molnupiravir Treatment on Patient-Reported COVID-19 Symptoms in the Phase 3 MOVe-OUT Trial: A Randomized, Placebo-Controlled Trial. Clin Infect Dis. 2023 Nov 30;77(11):1521-1530. doi: 10.1093/cid/ciad409. PMID 37466374
- [Derived] Chawla A, Birger R, Wan H, Cao Y, Maas BM, Paschke A, De Anda C, Rizk ML, Stone JA. Factors Influencing COVID-19 Risk: Insights From Molnupiravir Exposure-Response Modeling of Clinical Outcomes. Clin Pharmacol Ther. 2023 Jun;113(6):1337-1345. doi: 10.1002/cpt.2895. Epub 2023 Apr 27. PMID 37017631
- [Derived] Johnson MG, Strizki JM, Brown ML, Wan H, Shamsuddin HH, Ramgopal M, Florescu DF, Delobel P, Khaertynova I, Flores JF, Fouche LF, Chang SC, Williams-Diaz A, Du J, Grobler JA, Paschke A, De Anda C. Molnupiravir for the treatment of COVID-19 in immunocompromised participants: efficacy, safety, and virology results from the phase 3 randomized, placebo-controlled MOVe-OUT trial. Infection. 2023 Oct;51(5):1273-1284. doi: 10.1007/s15010-022-01959-9. Epub 2023 Jan 17. PMID 36648627
- [Derived] Johnson MG, Puenpatom A, Moncada PA, Burgess L, Duke ER, Ohmagari N, Wolf T, Bassetti M, Bhagani S, Ghosn J, Zhang Y, Wan H, Williams-Diaz A, Brown ML, Paschke A, De Anda C. Effect of Molnupiravir on Biomarkers, Respiratory Interventions, and Medical Services in COVID-19 : A Randomized, Placebo-Controlled Trial. Ann Intern Med. 2022 Aug;175(8):1126-1134. doi: 10.7326/M22-0729. Epub 2022 Jun 7. PMID 35667065
- [Derived] Jayk Bernal A, Gomes da Silva MM, Musungaie DB, Kovalchuk E, Gonzalez A, Delos Reyes V, Martin-Quiros A, Caraco Y, Williams-Diaz A, Brown ML, Du J, Pedley A, Assaid C, Strizki J, Grobler JA, Shamsuddin HH, Tipping R, Wan H, Paschke A, Butterton JR, Johnson MG, De Anda C; MOVe-OUT Study Group. Molnupiravir for Oral Treatment of Covid-19 in Nonhospitalized Patients. N Engl J Med. 2022 Feb 10;386(6):509-520. doi: 10.1056/NEJMoa2116044. Epub 2021 Dec 16. PMID 34914868

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 123 study centers in 21 countries.
Groups:
- Part 2: Molnupiravir 800 mg: 800 mg molnupiravir administered orally every 12 hours for 5 days (10 doses total)
Period: Overall Study
Arm/Group | Part 1: Molnupiravir 200 mg | Part 1: Molnupiravir 400 mg | Part 1: Molnupiravir 800 mg | Part 1: Placebo | Part 2: Molnupiravir 800 mg | Part 2: Placebo
Started | 75 | 77 | 76 | 74 | 716 | 717
Treated | 74 | 77 | 74 | 74 | 710 | 701
Completed | 71 | 74 | 71 | 69 | 675 | 663
Not Completed | 4 | 3 | 5 | 5 | 41 | 54
Not completed — Death | 0 | 0 | 0 | 1 | 3 | 14
Not completed — Lost to Follow-up | 2 | 1 | 1 | 2 | 10 | 8
Not completed — Withdrawal by Subject | 2 | 2 | 4 | 2 | 25 | 28
Not completed — Not Recorded | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Randomized By Mistake Without Study Treatment | 0 | 0 | 0 | 0 | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: Molnupiravir 200 mg | Part 1: Molnupiravir 400 mg | Part 1: Molnupiravir 800 mg | Part 1: Placebo | Part 2: Molnupiravir 800 mg | Part 2: Placebo | Total
Number analyzed (Participants) | 75 | 77 | 76 | 74 | 716 | 717 | 1735
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.5 (14.6) | 49.2 (14.2) | 51.0 (15.8) | 47.3 (15.2) | 44.4 (14.6) | 45.3 (15.0) | 45.6 (14.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 32 | 41 | 30 | 384 | 351 | 878
  Male | 35 | 45 | 35 | 44 | 332 | 366 | 857
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 29 | 30 | 23 | 33 | 355 | 356 | 826
  Not Hispanic or Latino | 46 | 46 | 51 | 39 | 355 | 358 | 895
  Unknown or Not Reported | 0 | 1 | 2 | 2 | 6 | 3 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 1 | 2 | 5 | 60 | 44 | 115
  Asian | 0 | 1 | 0 | 0 | 26 | 23 | 50
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 5 | 8 | 6 | 3 | 40 | 35 | 97
  White | 54 | 52 | 58 | 52 | 400 | 413 | 1029
  More than one race | 13 | 15 | 10 | 13 | 190 | 202 | 443
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 0 | 0 | 1
Time from Symptom Onset to Randomization (Part 1) [Count of Participants; unit: Participants] — Randomization of participants in Part 1 of this study was stratified by the time from symptom onset prior to the day of randomization (≤5 days or >5 days). Population: Analysis population consisted of all randomized participants in Part 1. Per protocol, this stratification factor was applicable to Part 1 of the study only.
  Participants
    ≤5 Days: number analyzed (Participants) | 75 | 77 | 76 | 74 | 0 | 0 | 302
    ≤5 Days | 51 | 52 | 52 | 50 |  |  | 205
    >5 Days: number analyzed (Participants) | 75 | 77 | 76 | 74 | 0 | 0 | 302
    >5 Days | 24 | 25 | 24 | 24 |  |  | 97
At Increased Risk of Severe Illness from Coronavirus Disease (COVID-19) (Part 1) [Count of Participants; unit: Participants] — Randomization of participants in Part 1 of this study was stratified by whether the participant was at an increased risk of severe illness from COVID-19 (Yes or No). Population: Analysis population consisted of all randomized participants in Part 1. Per protocol, this stratification factor was applicable to Part 1 of the study only.
  Participants
    Yes: number analyzed (Participants) | 75 | 77 | 76 | 74 | 0 | 0 | 302
    Yes | 56 | 58 | 57 | 56 |  |  | 227
    No: number analyzed (Participants) | 75 | 77 | 76 | 74 | 0 | 0 | 302
    No | 19 | 19 | 19 | 18 |  |  | 75
Time from Symptom Onset to Randomization (Part 2) [Count of Participants; unit: Participants] — Randomization of participants in Part 2 of this study was stratified by the time from symptom onset prior to the day of randomization (≤3 days or >3 days). Population: Analysis population consisted of all randomized participants in Part 2. Per protocol, this stratification factor was applicable to Part 2 of the study only.
  Participants
    ≤ 3 days: number analyzed (Participants) | 0 | 0 | 0 | 0 | 716 | 717 | 1433
    ≤ 3 days |  |  |  |  | 342 | 342 | 684
    > 3 days: number analyzed (Participants) | 0 | 0 | 0 | 0 | 716 | 717 | 1433
    > 3 days |  |  |  |  | 374 | 375 | 749

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Were Hospitalized and/or Died Through Day 29 (Primary Pre-specified Analysis)
Description: The percentage of participants who were hospitalized and/or died through Day 29 is presented. Hospitalization (all cause) is defined as at least 24 hours of acute care in a hospital or similar acute care facility. Death was due to any cause. Any participants with an unknown survival status at Day 29 were treated as failure. The analysis in Part 2 was based on all participants enrolled by the pre-specified futility/early efficacy analysis and was used for demonstration of superiority to placebo for the primary efficacy outcome measure.
Time Frame: Up to 29 days
Population: All randomized participants in Part 1 who received at least one dose of study intervention and were not hospitalized prior to the administration of the first dose of study intervention, and all randomized participants in Part 2 who had reached Day 29 by the pre-specified futility/early efficacy analysis who received at least one dose of study intervention and were not hospitalized prior to the administration of the first dose of study intervention, were analyzed.
Measure: Number; unit: Percentage of Participants
Arm/Group | Part 1: Molnupiravir 200 mg | Part 1: Molnupiravir 400 mg | Part 1: Molnupiravir 800 mg | Part 1: Placebo | Part 2: Molnupiravir 800 mg | Part 2: Placebo
Number analyzed (Participants) | 74 | 77 | 74 | 74 | 385 | 377
Percentage of Participants | 1.4 | 3.9 | 4.1 | 5.4 | 7.3 | 14.1
Statistical Analysis 1: Comparison: Part 1: Molnupiravir 200 mg vs Part 1: Placebo; Test type: Other — Difference in rates % and associated confidence intervals (CIs) were based on the Miettinen & Nurminen method stratified by randomization strata. Unknown survival status at Day 29 was treated as failure; Difference in Rates % = -4.1, 95% CI 2-sided [-12.2 to 2.5]
Statistical Analysis 2: Comparison: Part 1: Molnupiravir 400 mg vs Part 1: Placebo; Test type: Other — Difference in rates % and associated CIs were based on the Miettinen & Nurminen method stratified by randomization strata. Unknown survival status at Day 29 was treated as failure; Difference in Rates % = -1.5, 95% CI 2-sided [-9.9 to 6.2]
Statistical Analysis 3: Comparison: Part 1: Molnupiravir 800 mg vs Part 1: Placebo; Test type: Other — [test comment as in outcome 1, analysis 2]; Differences in Rates % = -1.3, 95% CI 2-sided [-9.6 to 6.4]
Statistical Analysis 4: Comparison: Part 2: Molnupiravir 800 mg vs Part 2: Placebo; Test type: Superiority — Difference in rates %, associated CIs, and p-value were based on the Miettinen & Nurminen method stratified by randomization strata. Unknown survival status at Day 29 was treated as failure; p = 0.0012, Miettinen & Nurminen; Difference in Rates % = -6.8, 95% CI 2-sided [-11.3 to -2.4]

2. Primary Outcome: Number of Participants With an Adverse Event (AE)
Description: The number of participants with at least 1 AE is presented. An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Time Frame: Up to 318 days
Population: All randomized participants who received at least one dose of study treatment were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Molnupiravir 200 mg | Part 1: Molnupiravir 400 mg | Part 1: Molnupiravir 800 mg | Part 1: Placebo | Part 2: Molnupiravir 800 mg | Part 2: Placebo
Number analyzed (Participants) | 74 | 77 | 74 | 74 | 710 | 701
Participants | 29 | 24 | 29 | 28 | 230 | 239

3. Primary Outcome: Number of Participants Who Discontinued Study Intervention Due to an AE
Description: The number of participants who discontinued study intervention due to an AE is presented. An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Time Frame: Up to 5 days
Population: All randomized participants who received at least one dose of study treatment were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Molnupiravir 200 mg | Part 1: Molnupiravir 400 mg | Part 1: Molnupiravir 800 mg | Part 1: Placebo | Part 2: Molnupiravir 800 mg | Part 2: Placebo
Number analyzed (Participants) | 74 | 77 | 74 | 74 | 710 | 701
Participants | 0 | 0 | 3 | 1 | 10 | 20

4. Secondary Outcome: Time to Sustained Resolution or Improvement of Each Targeted COVID-19 Sign/Symptom - Cough
Description: Time to sustained resolution or improvement of the targeted sign/symptom was defined as the number of days from randomization to the first of three consecutive days when resolution or improvement of the targeted sign/symptom was demonstrated and did not worsen by Day 29. The median number of days from randomization to the first day on or before study Day 29 for sustained resolution or improvement is presented. Per protocol, participants without the targeted sign/symptom reported at randomization were not included in the analysis.
Time Frame: Up to 29 days
Population: Per protocol, all randomized participants who received at least one dose of study intervention and had the corresponding sign or symptom (cough) at the time of randomization were analyzed.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Part 1: Molnupiravir 200 mg | Part 1: Molnupiravir 400 mg | Part 1: Molnupiravir 800 mg | Part 1: Placebo | Part 2: Molnupiravir 800 mg | Part 2: Placebo
Number analyzed (Participants) | 51 | 50 | 53 | 48 | 570 | 574
Days | 7.0 [5.0 to 10.0] | 6.5 [4.0 to 10.0] | 8.0 [6.0 to 11.0] | 6.0 [4.0 to 7.0] | 10.0 [9.0 to 11.0] | 10.0 [8.0 to 11.0]
Statistical Analysis 1: Comparison: Part 1: Molnupiravir 200 mg vs Part 1: Placebo; Test type: Other — Hazard ratio and associated CIs were based on Cox regression model with Efron's method of tie handling with treatment and randomization stratification factors as covariates; Hazard Ratio (HR) = 0.74, 95% CI 2-sided [0.48 to 1.13]
Statistical Analysis 2: Comparison: Part 1: Molnupiravir 400 mg vs Part 1: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 0.70, 95% CI 2-sided [0.46 to 1.08]
Statistical Analysis 3: Comparison: Part 1: Molnupiravir 800 mg vs Part 1: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 0.72, 95% CI 2-sided [0.47 to 1.11]
Statistical Analysis 4: Comparison: Part 2: Molnupiravir 800 mg vs Part 2: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 1.04, 95% CI 2-sided [0.92 to 1.18]

5. Secondary Outcome: Time to Sustained Resolution or Improvement of Each Targeted COVID-19 Sign/Symptom - Sore Throat
Description: as for outcome 4
Time Frame: Up to 29 days
Population: Per protocol, all randomized participants who received at least one dose of study intervention and had the corresponding sign or symptom (sore throat) at the time of randomization were analyzed.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Part 1: Molnupiravir 200 mg | Part 1: Molnupiravir 400 mg | Part 1: Molnupiravir 800 mg | Part 1: Placebo | Part 2: Molnupiravir 800 mg | Part 2: Placebo
Number analyzed (Participants) | 22 | 31 | 28 | 30 | 318 | 296
Days | 3.0 [2.0 to 4.0] | 3.0 [2.0 to 5.0] | 4.5 [3.0 to 8.0] | 5.0 [3.0 to 7.0] | 4.0 [4.0 to 5.0] | 5.0 [5.0 to 6.0]
Statistical Analysis 1: Comparison: Part 1: Molnupiravir 200 mg vs Part 1: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 1.49, 95% CI 2-sided [0.80 to 2.76]
Statistical Analysis 2: Comparison: Part 1: Molnupiravir 400 mg vs Part 1: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 1.20, 95% CI 2-sided [0.69 to 2.09]
Statistical Analysis 3: Comparison: Part 1: Molnupiravir 800 mg vs Part 1: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 0.93, 95% CI 2-sided [0.54 to 1.62]
Statistical Analysis 4: Comparison: Part 2: Molnupiravir 800 mg vs Part 2: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 1.12, 95% CI 2-sided [0.95 to 1.33]

6. Secondary Outcome: Time to Sustained Resolution or Improvement of Each Targeted COVID-19 Sign/Symptom - Nasal Congestion
Description: as for outcome 4
Time Frame: Up to 29 days
Population: Per protocol, all randomized participants who received at least one dose of study intervention and had the corresponding sign or symptom (nasal congestion) at the time of randomization were analyzed.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Part 1: Molnupiravir 200 mg | Part 1: Molnupiravir 400 mg | Part 1: Molnupiravir 800 mg | Part 1: Placebo | Part 2: Molnupiravir 800 mg | Part 2: Placebo
Number analyzed (Participants) | 48 | 41 | 40 | 54 | 439 | 429
Days | 4.0 [3.0 to 6.0] | 4.0 [3.0 to 7.0] | 8.0 [5.0 to 10.0] | 5.0 [4.0 to 6.0] | 5.0 [4.0 to 6.0] | 6.0 [5.0 to 7.0]
Statistical Analysis 1: Comparison: Part 1: Molnupiravir 200 mg vs Part 1: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 0.95, 95% CI 2-sided [0.62 to 1.46]
Statistical Analysis 2: Comparison: Part 1: Molnupiravir 400 mg vs Part 1: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 1.16, 95% CI 2-sided [0.75 to 1.79]
Statistical Analysis 3: Comparison: Part 1: Molnupiravir 800 mg vs Part 1: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 0.69, 95% CI 2-sided [0.45 to 1.07]
Statistical Analysis 4: Comparison: Part 2: Molnupiravir 800 mg vs Part 2: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 1.07, 95% CI 2-sided [0.93 to 1.23]

7. Secondary Outcome: Time to Sustained Resolution or Improvement of Each Targeted COVID-19 Sign/Symptom - Rhinorrhea
Description: as for outcome 4
Time Frame: Up to 29 days
Population: Per protocol, all randomized participants who received at least one dose of study intervention and had the corresponding sign or symptom (rhinorrhea) at the time of randomization were analyzed.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Part 1: Molnupiravir 200 mg | Part 1: Molnupiravir 400 mg | Part 1: Molnupiravir 800 mg | Part 1: Placebo | Part 2: Molnupiravir 800 mg | Part 2: Placebo
Number analyzed (Participants) | 31 | 30 | 17 | 35 | 348 | 347
Days | 4.0 [2.0 to 6.0] | 8.0 [5.0 to 10.0] | 9.0 [5.0 to 21.0] | 5.0 [3.0 to 6.0] | 5.0 [4.0 to 6.0] | 5.0 [5.0 to 6.0]
Statistical Analysis 1: Comparison: Part 1: Molnupiravir 200 mg vs Part 1: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 1.06, 95% CI 2-sided [0.62 to 1.83]
Statistical Analysis 2: Comparison: Part 1: Molnupiravir 400 mg vs Part 1: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 0.71, 95% CI 2-sided [0.40 to 1.26]
Statistical Analysis 3: Comparison: Part 1: Molnupiravir 800 mg vs Part 1: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 0.41, 95% CI 2-sided [0.20 to 0.85]
Statistical Analysis 4: Comparison: Part 2: Molnupiravir 800 mg vs Part 2: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 1.01, 95% CI 2-sided [0.86 to 1.18]

8. Secondary Outcome: Time to Sustained Resolution or Improvement of Each Targeted COVID-19 Sign/Symptom - Shortness of Breath or Difficulty Breathing
Description: as for outcome 4
Time Frame: Up to 29 days
Population: Per protocol, all randomized participants who received at least one dose of study intervention and had the corresponding sign or symptom (shortness of breath or difficulty breathing) at the time of randomization were analyzed.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Part 1: Molnupiravir 200 mg | Part 1: Molnupiravir 400 mg | Part 1: Molnupiravir 800 mg | Part 1: Placebo | Part 2: Molnupiravir 800 mg | Part 2: Placebo
Number analyzed (Participants) | 20 | 25 | 30 | 28 | 258 | 260
Days | 7.0 [4.0 to 22.0] | 4.0 [3.0 to 6.0] | 9.0 [4.0 to 17.0] | 5.0 [4.0 to 12.0] | 6.0 [6.0 to 8.0] | 9.0 [6.0 to 10.0]
Statistical Analysis 1: Comparison: Part 1: Molnupiravir 200 mg vs Part 1: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 0.66, 95% CI 2-sided [0.32 to 1.34]
Statistical Analysis 2: Comparison: Part 1: Molnupiravir 400 mg vs Part 1: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 1.44, 95% CI 2-sided [0.76 to 2.71]
Statistical Analysis 3: Comparison: Part 1: Molnupiravir 800 mg vs Part 1: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 0.75, 95% CI 2-sided [0.39 to 1.42]
Statistical Analysis 4: Comparison: Part 2: Molnupiravir 800 mg vs Part 2: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 1.14, 95% CI 2-sided [0.94 to 1.37]

9. Secondary Outcome: Time to Sustained Resolution or Improvement of Each Targeted COVID-19 Sign/Symptom - Muscles or Body Aches
Description: as for outcome 4
Time Frame: Up to 29 days
Population: Per protocol, all randomized participants who received at least one dose of study intervention and had the corresponding sign or symptom (muscles or body aches) at the time of randomization were analyzed.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Part 1: Molnupiravir 200 mg | Part 1: Molnupiravir 400 mg | Part 1: Molnupiravir 800 mg | Part 1: Placebo | Part 2: Molnupiravir 800 mg | Part 2: Placebo
Number analyzed (Participants) | 49 | 42 | 36 | 47 | 460 | 454
Days | 5.0 [3.0 to 7.0] | 4.0 [3.0 to 4.0] | 4.5 [3.0 to 15.0] | 4.0 [3.0 to 7.0] | 4.0 [4.0 to 5.0] | 5.0 [4.0 to 5.0]
Statistical Analysis 1: Comparison: Part 1: Molnupiravir 200 mg vs Part 1: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 1.03, 95% CI 2-sided [0.66 to 1.61]
Statistical Analysis 2: Comparison: Part 1: Molnupiravir 400 mg vs Part 1: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 1.32, 95% CI 2-sided [0.83 to 2.09]
Statistical Analysis 3: Comparison: Part 1: Molnupiravir 800 mg vs Part 1: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 0.76, 95% CI 2-sided [0.47 to 1.23]
Statistical Analysis 4: Comparison: Part 2: Molnupiravir 800 mg vs Part 2: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 1.01, 95% CI 2-sided [0.88 to 1.16]

10. Secondary Outcome: Time to Sustained Resolution or Improvement of Each Targeted COVID-19 Sign/Symptom - Fatigue
Description: as for outcome 4
Time Frame: Up to 29 days
Population: Per protocol, all randomized participants who received at least one dose of study intervention and had the corresponding sign or symptom (fatigue) at the time of randomization were analyzed.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Part 1: Molnupiravir 200 mg | Part 1: Molnupiravir 400 mg | Part 1: Molnupiravir 800 mg | Part 1: Placebo | Part 2: Molnupiravir 800 mg | Part 2: Placebo
Number analyzed (Participants) | 56 | 51 | 56 | 52 | 538 | 528
Days | 7.0 [4.0 to 11.0] | 5.0 [3.0 to 7.0] | 6.0 [4.0 to 11.0] | 6.0 [4.0 to 10.0] | 6.0 [6.0 to 7.0] | 7.0 [6.0 to 8.0]
Statistical Analysis 1: Comparison: Part 1: Molnupiravir 200 mg vs Part 1: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 0.93, 95% CI 2-sided [0.62 to 1.41]
Statistical Analysis 2: Comparison: Part 1: Molnupiravir 400 mg vs Part 1: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 1.09, 95% CI 2-sided [0.70 to 1.69]
Statistical Analysis 3: Comparison: Part 1: Molnupiravir 800 mg vs Part 1: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 1.00, 95% CI 2-sided [0.66 to 1.51]
Statistical Analysis 4: Comparison: Part 2: Molnupiravir 800 mg vs Part 2: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 1.15, 95% CI 2-sided [1.01 to 1.31]

11. Secondary Outcome: Time to Sustained Resolution or Improvement of Each Targeted COVID-19 Sign/Symptom - Feeling Hot or Feverish
Description: as for outcome 4
Time Frame: Up to 29 days
Population: Per protocol, all randomized participants who received at least one dose of study intervention and had the corresponding sign or symptom (feeling hot or feverish) at the time of randomization were analyzed.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Part 1: Molnupiravir 200 mg | Part 1: Molnupiravir 400 mg | Part 1: Molnupiravir 800 mg | Part 1: Placebo | Part 2: Molnupiravir 800 mg | Part 2: Placebo
Number analyzed (Participants) | 27 | 22 | 38 | 32 | 386 | 372
Days | 4.0 [3.0 to 6.0] | 2.0 [2.0 to 3.0] | 4.0 [3.0 to 5.0] | 3.5 [2.0 to 4.0] | 3.0 [3.0 to 4.0] | 4.0 [3.0 to 4.0]
Statistical Analysis 1: Comparison: Part 1: Molnupiravir 200 mg vs Part 1: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 0.96, 95% CI 2-sided [0.54 to 1.69]
Statistical Analysis 2: Comparison: Part 1: Molnupiravir 400 mg vs Part 1: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 1.10, 95% CI 2-sided [0.61 to 2.00]
Statistical Analysis 3: Comparison: Part 1: Molnupiravir 800 mg vs Part 1: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 0.83, 95% CI 2-sided [0.50 to 1.38]
Statistical Analysis 4: Comparison: Part 2: Molnupiravir 800 mg vs Part 2: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 1.04, 95% CI 2-sided [0.90 to 1.21]

12. Secondary Outcome: Time to Sustained Resolution or Improvement of Each Targeted COVID-19 Sign/Symptom - Chills
Description: as for outcome 4
Time Frame: Up to 29 days
Population: Per protocol, all randomized participants who received at least one dose of study intervention and had the corresponding sign or symptom (chills) at the time of randomization were analyzed.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Part 1: Molnupiravir 200 mg | Part 1: Molnupiravir 400 mg | Part 1: Molnupiravir 800 mg | Part 1: Placebo | Part 2: Molnupiravir 800 mg | Part 2: Placebo
Number analyzed (Participants) | 18 | 18 | 23 | 27 | 308 | 279
Days | 2.0 [2.0 to 5.0] | 2.0 [2.0 to 4.0] | 3.0 [2.0 to 3.0] | 4.0 [2.0 to 5.0] | 3.0 [2.0 to 3.0] | NA [NA to NA] — NA = Median time to resolution/improvement and upper and lower limits not reached due to insufficient number of participants with sustained resolution or improvement after randomization.
Statistical Analysis 1: Comparison: Part 1: Molnupiravir 200 mg vs Part 1: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 1.46, 95% CI 2-sided [0.77 to 2.76]
Statistical Analysis 2: Comparison: Part 1: Molnupiravir 400 mg vs Part 1: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 1.76, 95% CI 2-sided [0.92 to 3.38]
Statistical Analysis 3: Comparison: Part 1: Molnupiravir 800 mg vs Part 1: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 1.52, 95% CI 2-sided [0.81 to 2.86]
Statistical Analysis 4: Comparison: Part 2: Molnupiravir 800 mg vs Part 2: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 1.05, 95% CI 2-sided [0.89 to 1.24]

13. Secondary Outcome: Time to Sustained Resolution or Improvement of Each Targeted COVID-19 Sign/Symptom - Headache
Description: as for outcome 4
Time Frame: Up to 29 days
Population: Per protocol, all randomized participants who received at least one dose of study intervention and had the corresponding sign or symptom (headache) at the time of randomization were analyzed.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Part 1: Molnupiravir 200 mg | Part 1: Molnupiravir 400 mg | Part 1: Molnupiravir 800 mg | Part 1: Placebo | Part 2: Molnupiravir 800 mg | Part 2: Placebo
Number analyzed (Participants) | 39 | 42 | 35 | 37 | 472 | 429
Days | 4.0 [3.0 to 6.0] | 4.0 [3.0 to 7.0] | 4.0 [3.0 to 10.0] | 6.0 [3.0 to 10.0] | 5.0 [4.0 to 5.0] | 5.0 [5.0 to 6.0]
Statistical Analysis 1: Comparison: Part 1: Molnupiravir 200 mg vs Part 1: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 1.33, 95% CI 2-sided [0.81 to 2.20]
Statistical Analysis 2: Comparison: Part 1: Molnupiravir 400 mg vs Part 1: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 1.40, 95% CI 2-sided [0.85 to 2.31]
Statistical Analysis 3: Comparison: Part 1: Molnupiravir 800 mg vs Part 1: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 0.97, 95% CI 2-sided [0.57 to 1.65]
Statistical Analysis 4: Comparison: Part 2: Molnupiravir 800 mg vs Part 2: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 1.02, 95% CI 2-sided [0.89 to 1.18]

14. Secondary Outcome: Time to Sustained Resolution or Improvement of Each Targeted COVID-19 Sign/Symptom - Nausea
Description: as for outcome 4
Time Frame: Up to 29 days
Population: Per protocol, all randomized participants who received at least one dose of study intervention and had the corresponding sign or symptom (nausea) at the time of randomization were analyzed.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Part 1: Molnupiravir 200 mg | Part 1: Molnupiravir 400 mg | Part 1: Molnupiravir 800 mg | Part 1: Placebo | Part 2: Molnupiravir 800 mg | Part 2: Placebo
Number analyzed (Participants) | 16 | 17 | 10 | 16 | 176 | 171
Days | 5.0 [2.0 to 8.0] | 3.0 [2.0 to 4.0] | 6.0 [2.0 to 9.0] | 5.0 [2.0 to 9.0] | 4.0 [3.0 to 5.0] | 4.0 [3.0 to 4.0]
Statistical Analysis 1: Comparison: Part 1: Molnupiravir 200 mg vs Part 1: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 0.83, 95% CI 2-sided [0.36 to 1.91]
Statistical Analysis 2: Comparison: Part 1: Molnupiravir 400 mg vs Part 1: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 1.37, 95% CI 2-sided [0.64 to 2.97]
Statistical Analysis 3: Comparison: Part 1: Molnupiravir 800 mg vs Part 1: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 0.86, 95% CI 2-sided [0.37 to 2.02]
Statistical Analysis 4: Comparison: Part 2: Molnupiravir 800 mg vs Part 2: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 0.92, 95% CI 2-sided [0.74 to 1.14]

15. Secondary Outcome: Time to Sustained Resolution or Improvement of Each Targeted COVID-19 Sign/Symptom - Vomiting
Description: as for outcome 4
Time Frame: Up to 29 days
Population: Per protocol, all randomized participants who received at least one dose of study intervention and had the corresponding sign or symptom (vomiting) at the time of randomization were analyzed.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Part 1: Molnupiravir 200 mg | Part 1: Molnupiravir 400 mg | Part 1: Molnupiravir 800 mg | Part 1: Placebo | Part 2: Molnupiravir 800 mg | Part 2: Placebo
Number analyzed (Participants) | 2 | 2 | 2 | 5 | 49 | 38
Days | 4.0 [2.0 to 6.0] | 8.0 [2.0 to 14.0] | 5.0 [2.0 to 8.0] | 2.0 [2.0 to 4.0] | 3.0 [2.0 to 4.0] | NA [NA to NA] — NA = Median time to resolution/improvement and upper and lower limits not reached due to insufficient number of participants with sustained resolution or improvement after randomization.
Statistical Analysis 1: Comparison: Part 2: Molnupiravir 800 mg vs Part 2: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 0.68, 95% CI 2-sided [0.44 to 1.06]

16. Secondary Outcome: Time to Sustained Resolution or Improvement of Each Targeted COVID-19 Sign/Symptom - Diarrhea
Description: as for outcome 4
Time Frame: Up to 29 days
Population: Per protocol, all randomized participants who received at least one dose of study intervention and had the corresponding sign or symptom (diarrhea) at the time of randomization were analyzed.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Part 1: Molnupiravir 200 mg | Part 1: Molnupiravir 400 mg | Part 1: Molnupiravir 800 mg | Part 1: Placebo | Part 2: Molnupiravir 800 mg | Part 2: Placebo
Number analyzed (Participants) | 13 | 19 | 15 | 11 | 158 | 166
Days | 6.0 [2.0 to 13.0] | 4.0 [2.0 to 4.0] | 3.0 [2.0 to 6.0] | 2.0 [2.0 to 3.0] | 3.0 [3.0 to 4.0] | 3.0 [3.0 to 4.0]
Statistical Analysis 1: Comparison: Part 1: Molnupiravir 200 mg vs Part 1: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 0.21, 95% CI 2-sided [0.06 to 0.67]
Statistical Analysis 2: Comparison: Part 1: Molnupiravir 400 mg vs Part 1: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 0.33, 95% CI 2-sided [0.13 to 0.83]
Statistical Analysis 3: Comparison: Part 1: Molnupiravir 800 mg vs Part 1: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 0.27, 95% CI 2-sided [0.09 to 0.79]
Statistical Analysis 4: Comparison: Part 2: Molnupiravir 800 mg vs Part 2: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 1.09, 95% CI 2-sided [0.87 to 1.36]

17. Secondary Outcome: Time to Sustained Resolution or Improvement of Each Targeted COVID-19 Sign/Symptom - Loss of Taste
Description: as for outcome 4
Time Frame: Up to 29 days
Population: Per protocol, all randomized participants who received at least one dose of study intervention and had the corresponding sign or symptom (loss of taste) at the time of randomization were analyzed.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Part 1: Molnupiravir 200 mg | Part 1: Molnupiravir 400 mg | Part 1: Molnupiravir 800 mg | Part 1: Placebo | Part 2: Molnupiravir 800 mg | Part 2: Placebo
Number analyzed (Participants) | 33 | 15 | 18 | 30 | 242 | 262
Days | 6.0 [4.0 to 9.0] | 6.0 [4.0 to 11.0] | 10.0 [4.0 to 19.0] | 9.0 [5.0 to 16.0] | 9.0 [8.0 to 10.0] | 10.0 [8.0 to 12.0]
Statistical Analysis 1: Comparison: Part 1: Molnupiravir 200 mg vs Part 1: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 1.29, 95% CI 2-sided [0.74 to 2.23]
Statistical Analysis 2: Comparison: Part 1: Molnupiravir 400 mg vs Part 1: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 0.90, 95% CI 2-sided [0.45 to 1.80]
Statistical Analysis 3: Comparison: Part 1: Molnupiravir 800 mg vs Part 1: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 1.02, 95% CI 2-sided [0.55 to 1.89]
Statistical Analysis 4: Comparison: Part 2: Molnupiravir 800 mg vs Part 2: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 1.13, 95% CI 2-sided [0.94 to 1.37]

18. Secondary Outcome: Time to Sustained Resolution or Improvement of Each Targeted COVID-19 Sign/Symptom - Loss of Smell
Description: as for outcome 4
Time Frame: Up to 29 days
Population: Per protocol, all randomized participants who received at least one dose of study intervention and had the corresponding sign or symptom (loss of smell) at the time of randomization were analyzed.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Part 1: Molnupiravir 200 mg | Part 1: Molnupiravir 400 mg | Part 1: Molnupiravir 800 mg | Part 1: Placebo | Part 2: Molnupiravir 800 mg | Part 2: Placebo
Number analyzed (Participants) | 38 | 29 | 24 | 36 | 318 | 323
Days | 7.0 [6.0 to 9.0] | 10.0 [6.0 to 18.0] | 12.0 [6.0 to 19.0] | 12.0 [7.0 to 16.0] | 10.0 [9.0 to 11.0] | 11.0 [9.0 to 14.0]
Statistical Analysis 1: Comparison: Part 1: Molnupiravir 200 mg vs Part 1: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 1.39, 95% CI 2-sided [0.83 to 2.33]
Statistical Analysis 2: Comparison: Part 1: Molnupiravir 400 mg vs Part 1: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 0.86, 95% CI 2-sided [0.50 to 1.48]
Statistical Analysis 3: Comparison: Part 1: Molnupiravir 800 mg vs Part 1: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 0.98, 95% CI 2-sided [0.56 to 1.72]
Statistical Analysis 4: Comparison: Part 2: Molnupiravir 800 mg vs Part 2: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 1.20, 95% CI 2-sided [1.01 to 1.43]

19. Secondary Outcome: Time to Progression of Each Targeted COVID-19 Sign/Symptom - Cough
Description: Time to progression of the targeted sign/symptom was defined as the number of days from randomization to the first of two consecutive days when the targeted sign/symptom was worsened. The median number of days from randomization to the first day on or before study Day 29 for progression/worsening is presented. Per protocol, participants with symptoms reported at randomization as severe for the targeted sign/symptom were not included in the analysis.
Time Frame: Up to 29 days
Population: Per protocol, all randomized participants who received at least one dose of study intervention and reported absent or non-severe symptoms for the targeted sign/symptom (cough) at the time of randomization were analyzed.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Part 1: Molnupiravir 200 mg | Part 1: Molnupiravir 400 mg | Part 1: Molnupiravir 800 mg | Part 1: Placebo | Part 2: Molnupiravir 800 mg | Part 2: Placebo
Number analyzed (Participants) | 68 | 70 | 66 | 67 | 688 | 672
Days | NA [NA to NA] — NA = Median time to progression and upper and lower limits not reached due to an insufficient number of participants with progression after randomization. | NA [NA to NA] — NA = Median time to progression and upper and lower limits not reached due to an insufficient number of participants with progression after randomization. | NA [NA to NA] — NA = Median time to progression and upper and lower limits not reached due to an insufficient number of participants with progression after randomization. | NA [NA to NA] — NA = Median time to progression and upper and lower limits not reached due to an insufficient number of participants with progression after randomization. | NA [NA to NA] — NA = Median time to progression and upper and lower limits not reached due to an insufficient number of participants with progression after randomization. | NA [NA to NA] — NA = Median time to progression and upper and lower limits not reached due to an insufficient number of participants with progression after randomization.
Statistical Analysis 1: Comparison: Part 1: Molnupiravir 200 mg vs Part 1: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 0.79, 95% CI 2-sided [0.29 to 2.19]
Statistical Analysis 2: Comparison: Part 1: Molnupiravir 400 mg vs Part 1: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 0.91, 95% CI 2-sided [0.34 to 2.44]
Statistical Analysis 3: Comparison: Part 1: Molnupiravir 800 mg vs Part 1: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 1.77, 95% CI 2-sided [0.74 to 4.23]
Statistical Analysis 4: Comparison: Part 2: Molnupiravir 800 mg vs Part 2: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 0.83, 95% CI 2-sided [0.67 to 1.04]

20. Secondary Outcome: Time to Progression of Each Targeted COVID-19 Sign/Symptom - Sore Throat
Description: as for outcome 19
Time Frame: Up to 29 days
Population: Per protocol, all randomized participants who received at least one dose of study intervention and reported absent or non-severe symptoms for the targeted sign/symptom (sore throat) at the time of randomization were analyzed.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Part 1: Molnupiravir 200 mg | Part 1: Molnupiravir 400 mg | Part 1: Molnupiravir 800 mg | Part 1: Placebo | Part 2: Molnupiravir 800 mg | Part 2: Placebo
Number analyzed (Participants) | 71 | 72 | 70 | 67 | 695 | 681
Days | NA [NA to NA] — NA = Median time to progression and upper and lower limits not reached due to an insufficient number of participants with progression after randomization. | NA [NA to NA] — NA = Median time to progression and upper and lower limits not reached due to an insufficient number of participants with progression after randomization. | NA [NA to NA] — NA = Median time to progression and upper and lower limits not reached due to an insufficient number of participants with progression after randomization. | NA [NA to NA] — NA = Median time to progression and upper and lower limits not reached due to an insufficient number of participants with progression after randomization. | NA [NA to NA] — NA = Median time to progression and upper and lower limits not reached due to an insufficient number of participants with progression after randomization. | NA [NA to NA] — NA = Median time to progression and upper and lower limits not reached due to an insufficient number of participants with progression after randomization.
Statistical Analysis 1: Comparison: Part 1: Molnupiravir 200 mg vs Part 1: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 2.52, 95% CI 2-sided [0.98 to 6.53]
Statistical Analysis 2: Comparison: Part 1: Molnupiravir 400 mg vs Part 1: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 0.77, 95% CI 2-sided [0.23 to 2.52]
Statistical Analysis 3: Comparison: Part 1: Molnupiravir 800 mg vs Part 1: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 0.46, 95% CI 2-sided [0.11 to 1.84]
Statistical Analysis 4: Comparison: Part 2: Molnupiravir 800 mg vs Part 2: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 0.88, 95% CI 2-sided [0.66 to 1.16]

21. Secondary Outcome: Time to Progression of Each Targeted COVID-19 Sign/Symptom - Nasal Congestion
Description: as for outcome 19
Time Frame: Up to 29 days
Population: Per protocol, all randomized participants who received at least one dose of study intervention and reported absent or non-severe symptoms for the targeted sign/symptom (nasal congestion) at the time of randomization were analyzed.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Part 1: Molnupiravir 200 mg | Part 1: Molnupiravir 400 mg | Part 1: Molnupiravir 800 mg | Part 1: Placebo | Part 2: Molnupiravir 800 mg | Part 2: Placebo
Number analyzed (Participants) | 71 | 71 | 69 | 67 | 682 | 664
Days | NA [NA to NA] — NA = Median time to progression and upper and lower limits not reached due to an insufficient number of participants experiencing progression after randomization. | NA [NA to NA] — NA = Median time to progression and upper and lower limits not reached due to an insufficient number of participants experiencing progression after randomization. | NA [NA to NA] — NA = Median time to progression and upper and lower limits not reached due to an insufficient number of participants experiencing progression after randomization. | NA [NA to NA] — NA = Median time to progression and upper and lower limits not reached due to an insufficient number of participants experiencing progression after randomization. | NA [NA to NA] — NA = Median time to progression and upper and lower limits not reached due to an insufficient number of participants experiencing progression after randomization. | NA [NA to NA] — NA = Median time to progression and upper and lower limits not reached due to an insufficient number of participants experiencing progression after randomization.
Statistical Analysis 1: Comparison: Part 1: Molnupiravir 200 mg vs Part 1: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 1.23, 95% CI 2-sided [0.46 to 3.32]
Statistical Analysis 2: Comparison: Part 1: Molnupiravir 400 mg vs Part 1: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 1.42, 95% CI 2-sided [0.54 to 3.74]
Statistical Analysis 3: Comparison: Part 1: Molnupiravir 800 mg vs Part 1: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 0.97, 95% CI 2-sided [0.34 to 2.76]
Statistical Analysis 4: Comparison: Part 2: Molnupiravir 800 mg vs Part 2: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.66 to 1.10]

22. Secondary Outcome: Time to Progression of Each Targeted COVID-19 Sign/Symptom - Rhinorrhea
Description: as for outcome 19
Time Frame: Up to 29 days
Population: Per protocol, all randomized participants who received at least one dose of study intervention and reported absent or non-severe symptoms for the targeted sign/symptom (rhinorrhea) at the time of randomization were analyzed.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Part 1: Molnupiravir 200 mg | Part 1: Molnupiravir 400 mg | Part 1: Molnupiravir 800 mg | Part 1: Placebo | Part 2: Molnupiravir 800 mg | Part 2: Placebo
Number analyzed (Participants) | 71 | 72 | 65 | 67 | 694 | 690
Days | NA [NA to NA] — NA = Median time to progression and upper and lower limits not reached due to an insufficient number of participants with progression after randomization. | NA [NA to NA] — NA = Median time to progression and upper and lower limits not reached due to an insufficient number of participants with progression after randomization. | NA [NA to NA] — NA = Median time to progression and upper and lower limits not reached due to an insufficient number of participants with progression after randomization. | NA [NA to NA] — NA = Median time to progression and upper and lower limits not reached due to an insufficient number of participants with progression after randomization. | NA [NA to NA] — NA = Median time to progression and upper and lower limits not reached due to an insufficient number of participants with progression after randomization. | NA [NA to NA] — NA = Median time to progression and upper and lower limits not reached due to an insufficient number of participants with progression after randomization.
Statistical Analysis 1: Comparison: Part 1: Molnupiravir 200 mg vs Part 1: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 1.02, 95% CI 2-sided [0.41 to 2.52]
Statistical Analysis 2: Comparison: Part 1: Molnupiravir 400 mg vs Part 1: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 0.71, 95% CI 2-sided [0.26 to 1.90]
Statistical Analysis 3: Comparison: Part 1: Molnupiravir 800 mg vs Part 1: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 1.24, 95% CI 2-sided [0.51 to 3.00]
Statistical Analysis 4: Comparison: Part 2: Molnupiravir 800 mg vs Part 2: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 0.90, 95% CI 2-sided [0.69 to 1.17]

23. Secondary Outcome: Time to Progression of Each Targeted COVID-19 Sign/Symptom - Shortness of Breath or Difficulty Breathing
Description: as for outcome 19
Time Frame: Up to 29 days
Population: Per protocol, all randomized participants who received at least one dose of study intervention and reported absent or non-severe symptoms for the targeted sign/symptom (shortness of breath or difficulty breathing) at the time of randomization were analyzed.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Part 1: Molnupiravir 200 mg | Part 1: Molnupiravir 400 mg | Part 1: Molnupiravir 800 mg | Part 1: Placebo | Part 2: Molnupiravir 800 mg | Part 2: Placebo
Number analyzed (Participants) | 69 | 73 | 70 | 68 | 701 | 681
Days | NA [NA to NA] — NA = Median time to progression and upper and lower limits not reached due to an insufficient number of participants with progression after randomization. | NA [NA to NA] — NA = Median time to progression and upper and lower limits not reached due to an insufficient number of participants with progression after randomization. | NA [NA to NA] — NA = Median time to progression and upper and lower limits not reached due to an insufficient number of participants with progression after randomization. | NA [NA to NA] — NA = Median time to progression and upper and lower limits not reached due to an insufficient number of participants with progression after randomization. | NA [NA to NA] — NA = Median time to progression and upper and lower limits not reached due to an insufficient number of participants with progression after randomization. | NA [NA to NA] — NA = Median time to progression and upper and lower limits not reached due to an insufficient number of participants with progression after randomization.
Statistical Analysis 1: Comparison: Part 1: Molnupiravir 200 mg vs Part 1: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 0.80, 95% CI 2-sided [0.36 to 1.75]
Statistical Analysis 2: Comparison: Part 1: Molnupiravir 400 mg vs Part 1: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 0.73, 95% CI 2-sided [0.33 to 1.64]
Statistical Analysis 3: Comparison: Part 1: Molnupiravir 800 mg vs Part 1: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 0.71, 95% CI 2-sided [0.31 to 1.62]
Statistical Analysis 4: Comparison: Part 2: Molnupiravir 800 mg vs Part 2: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.76 to 1.16]

24. Secondary Outcome: Time to Progression of Each Targeted COVID-19 Sign/Symptom - Muscle or Body Aches
Description: as for outcome 19
Time Frame: Up to 29 days
Population: Per protocol, all randomized participants who received at least one dose of study intervention and reported absent or non-severe symptoms for the targeted sign/symptom (muscle or body aches) at the time of randomization were analyzed.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Part 1: Molnupiravir 200 mg | Part 1: Molnupiravir 400 mg | Part 1: Molnupiravir 800 mg | Part 1: Placebo | Part 2: Molnupiravir 800 mg | Part 2: Placebo
Number analyzed (Participants) | 66 | 71 | 68 | 62 | 655 | 640
Days | NA [NA to NA] — NA = Median time to progression and upper and lower limits not reached due to an insufficient number of participants with progression after randomization. | NA [NA to NA] — NA = Median time to progression and upper and lower limits not reached due to an insufficient number of participants with progression after randomization. | NA [NA to NA] — NA = Median time to progression and upper and lower limits not reached due to an insufficient number of participants with progression after randomization. | NA [NA to NA] — NA = Median time to progression and upper and lower limits not reached due to an insufficient number of participants with progression after randomization. | NA [NA to NA] — NA = Median time to progression and upper and lower limits not reached due to an insufficient number of participants with progression after randomization. | NA [NA to NA] — NA = Median time to progression and upper and lower limits not reached due to an insufficient number of participants with progression after randomization.
Statistical Analysis 1: Comparison: Part 1: Molnupiravir 200 mg vs Part 1: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 0.59, 95% CI 2-sided [0.25 to 1.39]
Statistical Analysis 2: Comparison: Part 1: Molnupiravir 400 mg vs Part 1: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 0.83, 95% CI 2-sided [0.38 to 1.78]
Statistical Analysis 3: Comparison: Part 1: Molnupiravir 800 mg vs Part 1: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 0.59, 95% CI 2-sided [0.25 to 1.39]
Statistical Analysis 4: Comparison: Part 2: Molnupiravir 800 mg vs Part 2: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 1.16, 95% CI 2-sided [0.91 to 1.48]

25. Secondary Outcome: Time to Progression of Each Targeted COVID-19 Sign/Symptom - Fatigue
Description: as for outcome 19
Time Frame: Up to 29 days
Population: Per protocol, all randomized participants who received at least one dose of study intervention and reported absent or non-severe symptoms for the targeted sign/symptom (fatigue) at the time of randomization were analyzed.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Part 1: Molnupiravir 200 mg | Part 1: Molnupiravir 400 mg | Part 1: Molnupiravir 800 mg | Part 1: Placebo | Part 2: Molnupiravir 800 mg | Part 2: Placebo
Number analyzed (Participants) | 64 | 69 | 62 | 60 | 659 | 637
Days | NA [NA to NA] — NA = Median time to progression and upper and lower limits not reached due to an insufficient number of participants with progression after randomization. | NA [NA to NA] — NA = Median time to progression and upper and lower limits not reached due to an insufficient number of participants with progression after randomization. | NA [NA to NA] — NA = Median time to progression and upper and lower limits not reached due to an insufficient number of participants with progression after randomization. | NA [NA to NA] — NA = Median time to progression and upper and lower limits not reached due to an insufficient number of participants with progression after randomization. | NA [NA to NA] — NA = Median time to progression and upper and lower limits not reached due to an insufficient number of participants with progression after randomization. | NA [NA to NA] — NA = Median time to progression and upper and lower limits not reached due to an insufficient number of participants with progression after randomization.
Statistical Analysis 1: Comparison: Part 1: Molnupiravir 200 mg vs Part 1: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 0.59, 95% CI 2-sided [0.26 to 1.34]
Statistical Analysis 2: Comparison: Part 1: Molnupiravir 400 mg vs Part 1: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 0.62, 95% CI 2-sided [0.28 to 1.37]
Statistical Analysis 3: Comparison: Part 1: Molnupiravir 800 mg vs Part 1: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 0.82, 95% CI 2-sided [0.38 to 1.74]
Statistical Analysis 4: Comparison: Part 2: Molnupiravir 800 mg vs Part 2: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 0.96, 95% CI 2-sided [0.79 to 1.21]

26. Secondary Outcome: Time to Progression of Each Targeted COVID-19 Sign/Symptom - Feeling Hot or Feverish
Description: as for outcome 19
Time Frame: Up to 29 days
Population: Per protocol, all randomized participants who received at least one dose of study intervention and reported absent or non-severe symptoms for the targeted sign/symptom (feeling hot or feverish) at the time of randomization were analyzed.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Part 1: Molnupiravir 200 mg | Part 1: Molnupiravir 400 mg | Part 1: Molnupiravir 800 mg | Part 1: Placebo | Part 2: Molnupiravir 800 mg | Part 2: Placebo
Number analyzed (Participants) | 68 | 71 | 65 | 66 | 676 | 673
Days | NA [NA to NA] — NA = Median time to progression and upper and lower limits not reached due to an insufficient number of participants with progression after randomization. | NA [NA to NA] — NA = Median time to progression and upper and lower limits not reached due to an insufficient number of participants with progression after randomization. | NA [NA to NA] — NA = Median time to progression and upper and lower limits not reached due to an insufficient number of participants with progression after randomization. | NA [NA to NA] — NA = Median time to progression and upper and lower limits not reached due to an insufficient number of participants with progression after randomization. | NA [NA to NA] — NA = Median time to progression and upper and lower limits not reached due to an insufficient number of participants with progression after randomization. | NA [NA to NA] — NA = Median time to progression and upper and lower limits not reached due to an insufficient number of participants with progression after randomization.
Statistical Analysis 1: Comparison: Part 1: Molnupiravir 200 mg vs Part 1: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 1.19, 95% CI 2-sided [0.47 to 3.02]
Statistical Analysis 2: Comparison: Part 1: Molnupiravir 400 mg vs Part 1: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 0.80, 95% CI 2-sided [0.29 to 2.20]
Statistical Analysis 3: Comparison: Part 1: Molnupiravir 800 mg vs Part 1: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 0.89, 95% CI 2-sided [0.32 to 2.45]
Statistical Analysis 4: Comparison: Part 2: Molnupiravir 800 mg vs Part 2: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 0.83, 95% CI 2-sided [0.62 to 1.11]

27. Secondary Outcome: Time to Progression of Each Targeted COVID-19 Sign/Symptom - Chills
Description: as for outcome 19
Time Frame: Up to 29 days
Population: Per protocol, all randomized participants who received at least one dose of study intervention and reported absent or non-severe symptoms for the targeted sign/symptom (chills) at the time of randomization were analyzed.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Part 1: Molnupiravir 200 mg | Part 1: Molnupiravir 400 mg | Part 1: Molnupiravir 800 mg | Part 1: Placebo | Part 2: Molnupiravir 800 mg | Part 2: Placebo
Number analyzed (Participants) | 68 | 72 | 70 | 66 | 679 | 676
Days | NA [NA to NA] — NA = Median time to progression and upper and lower limits not reached due to an insufficient number of participants with progression after randomization. | NA [NA to NA] — NA = Median time to progression and upper and lower limits not reached due to an insufficient number of participants with progression after randomization. | NA [NA to NA] — NA = Median time to progression and upper and lower limits not reached due to an insufficient number of participants with progression after randomization. | NA [NA to NA] — NA = Median time to progression and upper and lower limits not reached due to an insufficient number of participants with progression after randomization. | NA [NA to NA] — NA = Median time to progression and upper and lower limits not reached due to an insufficient number of participants with progression after randomization. | NA [NA to NA] — NA = Median time to progression and upper and lower limits not reached due to an insufficient number of participants with progression after randomization.
Statistical Analysis 1: Comparison: Part 1: Molnupiravir 200 mg vs Part 1: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 0.82, 95% CI 2-sided [0.30 to 2.27]
Statistical Analysis 2: Comparison: Part 1: Molnupiravir 400 mg vs Part 1: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 0.21, 95% CI 2-sided [0.04 to 1.00]
Statistical Analysis 3: Comparison: Part 1: Molnupiravir 800 mg vs Part 1: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 0.66, 95% CI 2-sided [0.23 to 1.91]
Statistical Analysis 4: Comparison: Part 2: Molnupiravir 800 mg vs Part 2: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 0.87, 95% CI 2-sided [0.62 to 1.23]

28. Secondary Outcome: Time to Progression of Each Targeted COVID-19 Sign/Symptom - Headache
Description: as for outcome 19
Time Frame: Up to 29 days
Population: Per protocol, all randomized participants who received at least one dose of study intervention and reported absent or non-severe symptoms for the targeted sign/symptom (headache) at the time of randomization were analyzed.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Part 1: Molnupiravir 200 mg | Part 1: Molnupiravir 400 mg | Part 1: Molnupiravir 800 mg | Part 1: Placebo | Part 2: Molnupiravir 800 mg | Part 2: Placebo
Number analyzed (Participants) | 69 | 72 | 69 | 67 | 640 | 640
Days | NA [NA to NA] — NA = Median time to progression and upper and lower limits not reached due to an insufficient number of participants with progression after randomization. | NA [NA to NA] — NA = Median time to progression and upper and lower limits not reached due to an insufficient number of participants with progression after randomization. | NA [NA to NA] — NA = Median time to progression and upper and lower limits not reached due to an insufficient number of participants with progression after randomization. | NA [NA to NA] — NA = Median time to progression and upper and lower limits not reached due to an insufficient number of participants with progression after randomization. | NA [NA to NA] — NA = Median time to progression and upper and lower limits not reached due to an insufficient number of participants with progression after randomization. | NA [NA to NA] — NA = Median time to progression and upper and lower limits not reached due to an insufficient number of participants with progression after randomization.
Statistical Analysis 1: Comparison: Part 1: Molnupiravir 200 mg vs Part 1: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 0.58, 95% CI 2-sided [0.28 to 1.20]
Statistical Analysis 2: Comparison: Part 1: Molnupiravir 400 mg vs Part 1: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 0.44, 95% CI 2-sided [0.20 to 0.95]
Statistical Analysis 3: Comparison: Part 1: Molnupiravir 800 mg vs Part 1: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 0.82, 95% CI 2-sided [0.43 to 1.59]
Statistical Analysis 4: Comparison: Part 2: Molnupiravir 800 mg vs Part 2: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 0.93, 95% CI 2-sided [0.73 to 1.19]

29. Secondary Outcome: Time to Progression of Each Targeted COVID-19 Sign/Symptom - Nausea
Description: as for outcome 19
Time Frame: Up to 29 days
Population: Per protocol, all randomized participants who received at least one dose of study intervention and reported absent or non-severe symptoms for the targeted sign/symptom (nausea) at the time of randomization were analyzed.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Part 1: Molnupiravir 200 mg | Part 1: Molnupiravir 400 mg | Part 1: Molnupiravir 800 mg | Part 1: Placebo | Part 2: Molnupiravir 800 mg | Part 2: Placebo
Number analyzed (Participants) | 72 | 73 | 70 | 69 | 688 | 686
Days | NA [NA to NA] — NA = Median time to progression and upper and lower limits not reached due to an insufficient number of participants with progression after randomization. | NA [NA to NA] — NA = Median time to progression and upper and lower limits not reached due to an insufficient number of participants with progression after randomization. | NA [NA to NA] — NA = Median time to progression and upper and lower limits not reached due to an insufficient number of participants with progression after randomization. | NA [NA to NA] — NA = Median time to progression and upper and lower limits not reached due to an insufficient number of participants with progression after randomization. | NA [NA to NA] — NA = Median time to progression and upper and lower limits not reached due to an insufficient number of participants with progression after randomization. | NA [NA to NA] — NA = Median time to progression and upper and lower limits not reached due to an insufficient number of participants with progression after randomization.
Statistical Analysis 1: Comparison: Part 1: Molnupiravir 200 mg vs Part 1: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 0.86, 95% CI 2-sided [0.35 to 2.11]
Statistical Analysis 2: Comparison: Part 1: Molnupiravir 400 mg vs Part 1: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 0.46, 95% CI 2-sided [0.16 to 1.34]
Statistical Analysis 3: Comparison: Part 1: Molnupiravir 800 mg vs Part 1: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 1.18, 95% CI 2-sided [0.50 to 2.79]
Statistical Analysis 4: Comparison: Part 2: Molnupiravir 800 mg vs Part 2: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 0.99, 95% CI 2-sided [0.74 to 1.32]

30. Secondary Outcome: Time to Progression of Each Targeted COVID-19 Sign/Symptom - Vomiting
Description: as for outcome 19
Time Frame: Up to 29 days
Population: Per protocol, all randomized participants who received at least one dose of study intervention and reported absent or non-severe symptoms for the targeted sign/symptom (vomiting) at the time of randomization were analyzed.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Part 1: Molnupiravir 200 mg | Part 1: Molnupiravir 400 mg | Part 1: Molnupiravir 800 mg | Part 1: Placebo | Part 2: Molnupiravir 800 mg | Part 2: Placebo
Number analyzed (Participants) | 72 | 73 | 71 | 69 | 702 | 692
Days | NA [NA to NA] — NA = Median time to progression and upper and lower limits not reached due to an insufficient number of participants with progression after randomization. | NA [NA to NA] — NA = Median time to progression and upper and lower limits not reached due to an insufficient number of participants with progression after randomization. | NA [NA to NA] — NA = Median time to progression and upper and lower limits not reached due to an insufficient number of participants with progression after randomization. | NA [NA to NA] — NA = Median time to progression and upper and lower limits not reached due to an insufficient number of participants with progression after randomization. | NA [NA to NA] — NA = Median time to progression and upper and lower limits not reached due to an insufficient number of participants with progression after randomization. | NA [NA to NA] — NA = Median time to progression and upper and lower limits not reached due to an insufficient number of participants with progression after randomization.
Statistical Analysis 1: Comparison: Part 1: Molnupiravir 200 mg vs Part 1: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 0.97, 95% CI 2-sided [0.06 to 15.54]
Statistical Analysis 2: Comparison: Part 1: Molnupiravir 400 mg vs Part 1: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 0.00, 95% CI 2-sided [lower limit 0.00] (NA = Upper limit not reached as no events were recorded)
Statistical Analysis 3: Comparison: Part 1: Molnupiravir 800 mg vs Part 1: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 1.00, 95% CI 2-sided [0.06 to 15.99]
Statistical Analysis 4: Comparison: Part 2: Molnupiravir 800 mg vs Part 2: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 0.76, 95% CI 2-sided [0.46 to 1.25]

31. Secondary Outcome: Time to Progression of Each Targeted COVID-19 Sign/Symptom - Diarrhea
Description: as for outcome 19
Time Frame: Up to 29 days
Population: Per protocol, all randomized participants who received at least one dose of study intervention and reported absent or non-severe symptoms for the targeted sign/symptom (diarrhea) at the time of randomization were analyzed.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Part 1: Molnupiravir 200 mg | Part 1: Molnupiravir 400 mg | Part 1: Molnupiravir 800 mg | Part 1: Placebo | Part 2: Molnupiravir 800 mg | Part 2: Placebo
Number analyzed (Participants) | 72 | 73 | 68 | 67 | 695 | 691
Days | NA [NA to NA] — NA = Median time to progression and upper and lower limits not reached due to an insufficient number of participants with progression after randomization. | NA [NA to NA] — NA = Median time to progression and upper and lower limits not reached due to an insufficient number of participants with progression after randomization. | NA [NA to NA] — NA = Median time to progression and upper and lower limits not reached due to an insufficient number of participants with progression after randomization. | NA [NA to NA] — NA = Median time to progression and upper and lower limits not reached due to an insufficient number of participants with progression after randomization. | NA [NA to NA] — NA = Median time to progression and upper and lower limits not reached due to an insufficient number of participants with progression after randomization. | NA [NA to NA] — NA = Median time to progression and upper and lower limits not reached due to an insufficient number of participants with progression after randomization.
Statistical Analysis 1: Comparison: Part 1: Molnupiravir 200 mg vs Part 1: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 1.49, 95% CI 2-sided [0.58 to 3.83]
Statistical Analysis 2: Comparison: Part 1: Molnupiravir 400 mg vs Part 1: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 1.14, 95% CI 2-sided [0.42 to 3.05]
Statistical Analysis 3: Comparison: Part 1: Molnupiravir 800 mg vs Part 1: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 1.49, 95% CI 2-sided [0.57 to 3.93]
Statistical Analysis 4: Comparison: Part 2: Molnupiravir 800 mg vs Part 2: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 0.82, 95% CI 2-sided [0.61 to 1.10]

32. Secondary Outcome: Time to Progression of Each Targeted COVID-19 Sign/Symptom - Loss of Taste
Description: as for outcome 19
Time Frame: Up to 29 days
Population: Per protocol, all randomized participants who received at least one dose of study intervention and reported absent or non-severe symptoms for the targeted sign/symptom (loss of taste) at the time of randomization were analyzed.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Part 1: Molnupiravir 200 mg | Part 1: Molnupiravir 400 mg | Part 1: Molnupiravir 800 mg | Part 1: Placebo | Part 2: Molnupiravir 800 mg | Part 2: Placebo
Number analyzed (Participants) | 38 | 56 | 48 | 37 | 461 | 433
Days | NA [NA to NA] — NA = Median time to progression and upper and lower limits not reached due to an insufficient number of participants with progression after randomization. | NA [NA to NA] — NA = Median time to progression and upper and lower limits not reached due to an insufficient number of participants with progression after randomization. | NA [NA to NA] — NA = Median time to progression and upper and lower limits not reached due to an insufficient number of participants with progression after randomization. | NA [NA to NA] — NA = Median time to progression and upper and lower limits not reached due to an insufficient number of participants with progression after randomization. | NA [NA to NA] — NA = Median time to progression and upper and lower limits not reached due to an insufficient number of participants with progression after randomization. | NA [NA to NA] — NA = Median time to progression and upper and lower limits not reached due to an insufficient number of participants with progression after randomization.
Statistical Analysis 1: Comparison: Part 1: Molnupiravir 200 mg vs Part 1: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 0.36, 95% CI 2-sided [0.11 to 1.21]
Statistical Analysis 2: Comparison: Part 1: Molnupiravir 400 mg vs Part 1: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 0.52, 95% CI 2-sided [0.20 to 1.36]
Statistical Analysis 3: Comparison: Part 1: Molnupiravir 800 mg vs Part 1: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 0.74, 95% CI 2-sided [0.29 to 1.89]
Statistical Analysis 4: Comparison: Part 2: Molnupiravir 800 mg vs Part 2: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 0.91, 95% CI 2-sided [0.68 to 1.20]

33. Secondary Outcome: Time to Progression of Each Targeted COVID-19 Sign/Symptom - Loss of Smell
Description: as for outcome 19
Time Frame: Up to 29 days
Population: Per protocol, all randomized participants who received at least one dose of study intervention and reported absent or non-severe symptoms for the targeted sign/symptom (loss of smell) at the time of randomization were analyzed.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Part 1: Molnupiravir 200 mg | Part 1: Molnupiravir 400 mg | Part 1: Molnupiravir 800 mg | Part 1: Placebo | Part 2: Molnupiravir 800 mg | Part 2: Placebo
Number analyzed (Participants) | 33 | 42 | 42 | 31 | 385 | 372
Days | NA [NA to NA] — NA = Median time to progression and upper and lower limits not reached due to an insufficient number of participants with progression after randomization. | NA [NA to NA] — NA = Median time to progression and upper and lower limits not reached due to an insufficient number of participants with progression after randomization. | NA [NA to NA] — NA = Median time to progression and upper and lower limits not reached due to an insufficient number of participants with progression after randomization. | NA [NA to NA] — NA = Median time to progression and upper and lower limits not reached due to an insufficient number of participants with progression after randomization. | NA [NA to NA] — NA = Median time to progression and upper and lower limits not reached due to an insufficient number of participants with progression after randomization. | NA [NA to NA] — NA = Median time to progression and upper and lower limits not reached due to an insufficient number of participants with progression after randomization.
Statistical Analysis 1: Comparison: Part 1: Molnupiravir 200 mg vs Part 1: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 0.35, 95% CI 2-sided [0.09 to 1.33]
Statistical Analysis 2: Comparison: Part 1: Molnupiravir 400 mg vs Part 1: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 0.80, 95% CI 2-sided [0.30 to 2.15]
Statistical Analysis 3: Comparison: Part 1: Molnupiravir 800 mg vs Part 1: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 0.51, 95% CI 2-sided [0.18 to 1.48]
Statistical Analysis 4: Comparison: Part 2: Molnupiravir 800 mg vs Part 2: Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 0.81, 95% CI 2-sided [0.62 to 1.04]

34. Secondary Outcome: Number of Participants With Responses on WHO 11-point Ordinal Outcomes Score on a Scale on Day 3
Description: The World Health Organization (WHO) outcome scale is an 11-point ordinal score that categorizes clinical progression. Score ranges from 0 ("uninfected") to 10 ("dead") with higher score indicating clinical progression. The number of participants at each score category is presented.
Time Frame: Day 3
Population: Per protocol, all randomized participants who received at least one dose of study treatment and had non-missing ordinal scale data at the time point assessed were analyzed. 38 participants with missing ordinal scale data were not included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Molnupiravir 200 mg | Part 1: Molnupiravir 400 mg | Part 1: Molnupiravir 800 mg | Part 1: Placebo | Part 2: Molnupiravir 800 mg | Part 2: Placebo
Number analyzed (Participants) | 72 | 75 | 73 | 70 | 695 | 684
Participants
  0 | 2 | 0 | 0 | 1 | 2 | 3
  1 | 2 | 2 | 1 | 1 | 11 | 13
  2 | 68 | 72 | 66 | 66 | 655 | 640
  3 | 0 | 0 | 2 | 2 | 13 | 10
  4 | 0 | 1 | 3 | 0 | 7 | 4
  5 | 0 | 0 | 1 | 0 | 4 | 13
  6 | 0 | 0 | 0 | 0 | 3 | 1
  7 | 0 | 0 | 0 | 0 | 0 | 0
  8 | 0 | 0 | 0 | 0 | 0 | 0
  9 | 0 | 0 | 0 | 0 | 0 | 0
  10 | 0 | 0 | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: Part 1: Molnupiravir 200 mg vs Part 1: Placebo; Test type: Other — Odds ratio was based on the proportional odds model with WHO-11 score categories as the response variable. Due to sparse data, the final model includes only treatment as covariate. CIs are based on Wald Chi-Square Test; Odds Ratio (OR) = 3.04, 95% CI 2-sided [0.59 to 15.59]
Statistical Analysis 2: Comparison: Part 1: Molnupiravir 400 mg vs Part 1: Placebo; Test type: Other — [test comment as in outcome 34, analysis 1]; Odds Ratio (OR) = 1.33, 95% CI 2-sided [0.29 to 6.16]
Statistical Analysis 3: Comparison: Part 1: Molnupiravir 800 mg vs Part 1: Placebo; Test type: Other — [test comment as in outcome 34, analysis 1]; Odds Ratio (OR) = 0.37, 95% CI 2-sided [0.09 to 1.44]
Statistical Analysis 4: Comparison: Part 2: Molnupiravir 800 mg vs Part 2: Placebo; Test type: Other — [test comment as in outcome 34, analysis 1]; Odds Ratio (OR) = 1.19, 95% CI 2-sided [0.62 to 2.30]

35. Secondary Outcome: Number of Participants With Responses on WHO 11-point Ordinal Outcomes Score on a Scale on End of Treatment (EOT [Day 5])
Description: as for outcome 34
Time Frame: EOT (Day 5)
Population: Per protocol, all randomized participants who received at least one dose of study treatment and had non-missing ordinal scale data at the time point assessed were analyzed. 40 participants with missing ordinal scale data were not included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Molnupiravir 200 mg | Part 1: Molnupiravir 400 mg | Part 1: Molnupiravir 800 mg | Part 1: Placebo | Part 2: Molnupiravir 800 mg | Part 2: Placebo
Number analyzed (Participants) | 70 | 75 | 71 | 70 | 697 | 684
Participants
  0 | 3 | 0 | 2 | 1 | 11 | 10
  1 | 9 | 5 | 3 | 3 | 36 | 34
  2 | 58 | 69 | 63 | 65 | 613 | 593
  3 | 0 | 0 | 0 | 1 | 14 | 9
  4 | 0 | 0 | 1 | 0 | 10 | 13
  5 | 0 | 1 | 1 | 0 | 7 | 21
  6 | 0 | 0 | 0 | 0 | 5 | 2
  7 | 0 | 0 | 0 | 0 | 0 | 1
  8 | 0 | 0 | 1 | 0 | 0 | 1
  9 | 0 | 0 | 0 | 0 | 1 | 0
  10 | 0 | 0 | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: Part 1: Molnupiravir 200 mg vs Part 1: Placebo; Test type: Other — [test comment as in outcome 34, analysis 1]; Odds Ratio (OR) = 3.67, 95% CI 2-sided [1.14 to 11.88]
Statistical Analysis 2: Comparison: Part 1: Molnupiravir 400 mg vs Part 1: Placebo; Test type: Other — [test comment as in outcome 34, analysis 1]; Odds Ratio (OR) = 1.16, 95% CI 2-sided [0.34 to 3.98]
Statistical Analysis 3: Comparison: Part 1: Molnupiravir 800 mg vs Part 1: Placebo; Test type: Other — [test comment as in outcome 34, analysis 1]; Odds Ratio (OR) = 0.85, 95% CI 2-sided [0.27 to 2.68]
Statistical Analysis 4: Comparison: Part 2: Molnupiravir 800 mg vs Part 2: Placebo; Test type: Other — [test comment as in outcome 34, analysis 1]; Odds Ratio (OR) = 1.52, 95% CI 2-sided [0.96 to 2.39]

36. Secondary Outcome: Number of Participants With Responses on WHO 11-point Ordinal Outcomes Score on a Scale on Day 10
Description: as for outcome 34
Time Frame: Day 10
Population: Per protocol, all randomized participants who received at least one dose of study treatment and had non-missing ordinal scale data at the time point assessed were analyzed. 80 participants with missing ordinal scale data were not included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Molnupiravir 200 mg | Part 1: Molnupiravir 400 mg | Part 1: Molnupiravir 800 mg | Part 1: Placebo | Part 2: Molnupiravir 800 mg | Part 2: Placebo
Number analyzed (Participants) | 70 | 73 | 69 | 69 | 673 | 673
Participants
  0 | 9 | 11 | 3 | 4 | 40 | 32
  1 | 15 | 8 | 7 | 13 | 68 | 81
  2 | 45 | 52 | 56 | 49 | 519 | 493
  3 | 0 | 0 | 0 | 0 | 12 | 6
  4 | 0 | 0 | 1 | 2 | 16 | 23
  5 | 1 | 1 | 1 | 1 | 11 | 21
  6 | 0 | 1 | 0 | 0 | 4 | 11
  7 | 0 | 0 | 0 | 0 | 1 | 2
  8 | 0 | 0 | 1 | 0 | 2 | 3
  9 | 0 | 0 | 0 | 0 | 0 | 1
  10 | 0 | 0 | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: Part 1: Molnupiravir 200 mg vs Part 1: Placebo; Test type: Other — [test comment as in outcome 34, analysis 1]; Odds Ratio (OR) = 1.68, 95% CI 2-sided [0.82 to 3.45]
Statistical Analysis 2: Comparison: Part 1: Molnupiravir 400 mg vs Part 1: Placebo; Test type: Other — [test comment as in outcome 34, analysis 1]; Odds Ratio (OR) = 1.13, 95% CI 2-sided [0.55 to 2.33]
Statistical Analysis 3: Comparison: Part 1: Molnupiravir 800 mg vs Part 1: Placebo; Test type: Other — [test comment as in outcome 34, analysis 1]; Odds Ratio (OR) = 0.59, 95% CI 2-sided [0.27 to 1.29]
Statistical Analysis 4: Comparison: Part 2: Molnupiravir 800 mg vs Part 2: Placebo; Test type: Other — [test comment as in outcome 34, analysis 1]; Odds Ratio (OR) = 1.58, 95% CI 2-sided [1.14 to 2.20]

37. Secondary Outcome: Number of Participants With Responses on WHO 11-point Ordinal Outcomes Score on a Scale on Day 15
Description: as for outcome 34
Time Frame: Day 15
Population: Per protocol, all randomized participants who received at least one dose of study treatment and had non-missing ordinal scale data at the time point assessed were analyzed. 87 participants with missing ordinal scale data were not included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Molnupiravir 200 mg | Part 1: Molnupiravir 400 mg | Part 1: Molnupiravir 800 mg | Part 1: Placebo | Part 2: Molnupiravir 800 mg | Part 2: Placebo
Number analyzed (Participants) | 72 | 73 | 70 | 69 | 669 | 667
Participants
  0 | 20 | 21 | 13 | 11 | 102 | 94
  1 | 15 | 8 | 9 | 17 | 110 | 92
  2 | 36 | 43 | 45 | 39 | 433 | 427
  3 | 0 | 0 | 0 | 0 | 5 | 6
  4 | 1 | 0 | 1 | 2 | 11 | 21
  5 | 0 | 0 | 1 | 0 | 4 | 12
  6 | 0 | 1 | 0 | 0 | 1 | 6
  7 | 0 | 0 | 0 | 0 | 1 | 2
  8 | 0 | 0 | 1 | 0 | 2 | 2
  9 | 0 | 0 | 0 | 0 | 0 | 0
  10 | 0 | 0 | 0 | 0 | 0 | 5
Statistical Analysis 1: Comparison: Part 1: Molnupiravir 200 mg vs Part 1: Placebo; Test type: Other — [test comment as in outcome 34, analysis 1]; Odds Ratio (OR) = 1.41, 95% CI 2-sided [0.73 to 2.73]
Statistical Analysis 2: Comparison: Part 1: Molnupiravir 400 mg vs Part 1: Placebo; Test type: Other — [test comment as in outcome 34, analysis 1]; Odds Ratio (OR) = 1.00, 95% CI 2-sided [0.52 to 1.94]
Statistical Analysis 3: Comparison: Part 1: Molnupiravir 800 mg vs Part 1: Placebo; Test type: Other — [test comment as in outcome 34, analysis 1]; Odds Ratio (OR) = 0.67, 95% CI 2-sided [0.34 to 1.32]
Statistical Analysis 4: Comparison: Part 2: Molnupiravir 800 mg vs Part 2: Placebo; Test type: Other — [test comment as in outcome 34, analysis 1]; Odds Ratio (OR) = 1.36, 95% CI 2-sided [1.03 to 1.78]

38. Secondary Outcome: Number of Participants With Responses on WHO 11-point Ordinal Outcomes Score on a Scale on Day 29
Description: as for outcome 34
Time Frame: Day 29
Population: Per protocol, all randomized participants who received at least one dose of study treatment and had non-missing ordinal scale data at the time point assessed were analyzed. 139 participants with missing ordinal scale data were not included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Molnupiravir 200 mg | Part 1: Molnupiravir 400 mg | Part 1: Molnupiravir 800 mg | Part 1: Placebo | Part 2: Molnupiravir 800 mg | Part 2: Placebo
Number analyzed (Participants) | 68 | 72 | 66 | 67 | 645 | 650
Participants
  0 | 35 | 40 | 39 | 36 | 312 | 314
  1 | 14 | 13 | 10 | 16 | 126 | 115
  2 | 19 | 19 | 15 | 14 | 197 | 198
  3 | 0 | 0 | 0 | 0 | 1 | 1
  4 | 0 | 0 | 2 | 1 | 4 | 10
  5 | 0 | 0 | 0 | 0 | 2 | 2
  6 | 0 | 0 | 0 | 0 | 0 | 0
  7 | 0 | 0 | 0 | 0 | 0 | 1
  8 | 0 | 0 | 0 | 0 | 2 | 0
  9 | 0 | 0 | 0 | 0 | 0 | 0
  10 | 0 | 0 | 0 | 0 | 1 | 9
Statistical Analysis 1: Comparison: Part 1: Molnupiravir 200 mg vs Part 1: Placebo; Test type: Other — [test comment as in outcome 34, analysis 1]; Odds Ratio (OR) = 0.76, 95% CI 2-sided [0.35 to 1.66]
Statistical Analysis 2: Comparison: Part 1: Molnupiravir 400 mg vs Part 1: Placebo; Test type: Other — [test comment as in outcome 34, analysis 1]; Odds Ratio (OR) = 0.82, 95% CI 2-sided [0.38 to 1.79]
Statistical Analysis 3: Comparison: Part 1: Molnupiravir 800 mg vs Part 1: Placebo; Test type: Other — [test comment as in outcome 34, analysis 1]; Odds Ratio (OR) = 0.82, 95% CI 2-sided [0.37 to 1.81]
Statistical Analysis 4: Comparison: Part 2: Molnupiravir 800 mg vs Part 2: Placebo; Test type: Other — [test comment as in outcome 34, analysis 1]; Odds Ratio (OR) = 1.04, 95% CI 2-sided [0.84 to 1.29]

39. Post Hoc Outcome: Percentage of Participants Who Were Hospitalized and/or Died Through Day 29
Description: The percentage of participants who were hospitalized and/or died through Day 29 is presented. Hospitalization (all cause) is defined as at least 24 hours of acute care in a hospital or similar acute care facility. Death was due to any cause. Any participants with an unknown survival status at Day 29 were treated as failure. This analysis was based on all randomized participants in Part 2 who received at least one dose of study treatment, were not hospitalized prior to the administration of the first dose of study intervention, and had reached Day 29 post treatment.
Time Frame: Up to 29 days
Population: All randomized participants in Part 2 who received at least one dose of study intervention and were not hospitalized prior to the administration of the first dose of study intervention were analyzed.
Measure: Number; unit: Percentage of Participants
Arm/Group | Part 2: Molnupiravir 800 mg | Part 2: Placebo
Number analyzed (Participants) | 709 | 699
Percentage of Participants | 6.8 | 9.7
Statistical Analysis 1: Comparison: Part 2: Molnupiravir 800 mg vs Part 2: Placebo; Test type: Other — [test comment as in outcome 1, analysis 2]; Difference in Rates % = -3.0, 95% CI 2-sided [-5.9 to -0.1]

ADVERSE EVENTS:
Time Frame: Up to 318 days
Description: The analysis population for All-Cause Mortality included all randomized participants. The safety analysis population included all randomized participants who received at least one dose of study treatment.
Groups:
- Part 1: MK-4482 200 mg: 200 mg molnupiravir administered orally every 12 hours for 5 days (10 doses total)
- Part 1: MK-4482 400 mg: 400 mg molnupiravir administered orally every 12 hours for 5 days (10 doses total)
- Part 1: MK-4482 800 mg; Part 2: MK-4482 800 mg: 800 mg molnupiravir administered orally every 12 hours for 5 days (10 doses total)
Arm/Group | Part 1: MK-4482 200 mg | Part 1: MK-4482 400 mg | Part 1: MK-4482 800 mg | Part 1: Placebo | Part 2: MK-4482 800 mg | Part 2: Placebo
All-Cause Mortality (participants affected / at risk) | 0/75 | 0/77 | 0/76 | 1/74 | 4/716 | 16/717
Serious Adverse Events (participants affected / at risk) | 1/74 | 3/77 | 4/74 | 5/74 | 51/710 | 67/701
Other Adverse Events (participants affected / at risk) | 6/74 | 4/77 | 5/74 | 9/74 | 38/710 | 38/701
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: MK-4482 200 mg (N=74) | Part 1: MK-4482 400 mg (N=77) | Part 1: MK-4482 800 mg (N=74) | Part 1: Placebo (N=74) | Part 2: MK-4482 800 mg (N=710) | Part 2: Placebo (N=701)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 37 (37) | 53 (53)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 2 (2) | 2 (2) | 2 (2) | 29 (29) | 43 (43)
Lung abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peritonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Pneumonia aspiration (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
Pneumonia haemophilus (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 9 (9)
Peripheral vascular disorder (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Shock (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thrombosis mesenteric vessel (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia staphylococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: MK-4482 200 mg (N=74) | Part 1: MK-4482 400 mg (N=77) | Part 1: MK-4482 800 mg (N=74) | Part 1: Placebo (N=74) | Part 2: MK-4482 800 mg (N=710) | Part 2: Placebo (N=701)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 2 (2) | 2 (2) | 4 (5) | 16 (17) | 21 (22)
COVID-19 (Infections and infestations) | 3 (3) | 2 (2) | 3 (3) | 5 (5) | 23 (24) | 17 (17)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor will generally support publication of multicenter studies only in their entirety and not as individual site data. In this case, a coordinating investigator will be designated by mutual agreement. If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-15): https://cdn.clinicaltrials.gov/large-docs/97/NCT04575597/Prot_SAP_000.pdf